# Reporting and Analysis Plan

**Study ID: 207804** 

**Official Title of Study:** Reporting and Analysis Plan for study 207804 A two-part phase I randomized, double-blind, placebo-controlled study toevaluate safety, tolerability, pharmacokinetics and target engagement of single intravenous and subcutaneous doses of GSK3858279 in healthy participants and to evaluate the efficacy of repeat subcutaneous doses in participants with osteoarthritis of the knee

NCT Number: NCT03485365

Date of Document: 28-JUL-2022

#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | Ξ | Reporting and Analysis Plan for Study 207804: A two-part phase I randomized, double-blind, placebo-controlled study to evaluate safety, tolerability, pharmacokinetics and target engagement of single intravenous and subcutaneous doses of GSK3858279 in healthy participants and to evaluate the efficacy of repeat subcutaneous doses in participants with osteoarthritis of the knee |
|---|---|---|
| Compound Number | : | GSK3858279 |
| Study Number | : | 207804 |
| Effective Date | : | 28-JUL-2022 |

#### Description:

The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report from Part A and Part B of Protocol 207804.

This RAP is intended to evaluate the:

- safety, tolerability, pharmacokinetics and target engagement of GSK3858279 in single intravenous and subcutaneous doses in healthy participants (Part A)
- safety, tolerability, efficacy, pharmacokinetics, target engagement and immunogenicity of repeat subcutaneous doses in participants with osteoarthritis of the knee (Part B).

This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverables.

| Author | Date |
|--------------------|-------------|
| PPD | |
| Study Statistician | 28-JUL-2022 |
| PPD | |
| CPMS Study Lead | |

Copyright 2022 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited

# **RAP Team Review Confirmations**

(Method: E-mail)

| Reviewer | Date |
|-------------------------------------------|------------|
| Clinical Science Lead and Medical Monitor | 11-ЛП-2022 |
| CPMS Project Lead | |
| Global Safety Representative 12-JUL-2022 | |

# Clinical Statistics Line Approvals

(Method: eSignature/email)

| Approver | Date |
|----------------------------|-------------|
| Project Statistician | 21-JUL-2022 |
| Project Programming Leader | 28-JUL-2022 |

# **TABLE OF CONTENTS**

| 1. | | |
|---|---|---|
| | 1.1. Version history | 6 |
| 2. | SUMMARY OF KEY PROTOCOL INFORMATION | 7 |
| | 2.1. Changes to the Protocol Defined Statistical Analysis Plan | 7 |
| | 2.2. Study Objectives and Endpoints | |
| | 2.3. Study Design | |
| | 2.4. Statistical Analyses | |
| 3. | PLANNED ANALYSES | 13 |
| ٥. | 3.1. Interim Analyses | |
| | 3.2. Final Analyses | |
| 4 | ANALYSIS POPULATIONS | 15 |
| ٦. | 4.1. Analysis Populations | |
| | 4.1.1. Part A and B | |
| | 4.1.2. Part A only | |
| | , | |
| | 4.1.3. Part B only | |
| | 4.2. Flotocol Deviations | 10 |
| <b>5</b> . | | |
| | CONVENTIONS | 18 |
| | 5.1. General | |
| | 5.2. Study Treatment Display Descriptors | |
| | 5.3. Baseline Definitions | 18 |
| | 5.4. Other Considerations for Data Analyses and Data Handling | |
| | Conventions | 19 |
| 6. | STUDY POPULATION ANALYSES | 20 |
| 7. | EFFICACY ANALYSES – PART B ONLY | 21 |
| • | 7.1. Co-primary Efficacy Analyses | |
| | 7.1.1. Endpoint / Variables | |
| | 7.1.2. Summary Measure | |
| | 7.1.3. Population of Interest | |
| | 7.1.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | 7.1.5. Statistical Analyses / Methods | |
| | 7.2. Exploratory Efficacy Analyses | |
| | CCI | |
| | 7.2.2. Summary Measure | |
| | 7.2.3. Population of Interest | |
| | <ol> <li>7.2.4. Strategy for Intercurrent (Post-Randomization) Events</li> </ol> | |
| | 7.2.5. Statistical Analyses / Methods | 25 |
| 8. | SAFETY ANALYSES | 26 |
| | 8.1. Adverse Events Analyses | |
| | 8.2. Clinical Laboratory Analyses | |
| | 8.3. Other Safety Analyses | |
| | 8.4. COVID-19 Pandemic Statistical Displays | |
| 9. | PHARMACOKINETIC ANALYSES | 20 |
| J. | I HARMAOORINE HO AMALTOES | |


| | 9.1. | Serum Pharmacokinetics | 30 |
|---|---|---|---|
| | | 9.1.1. Endpoint / Variables | 30 |
| | | 9.1.2. Summary Measure | 32 |
| | | 9.1.3. Population of Interest | 32 |
| | | 9.1.4. Strategy for Intercurrent (Post-Randomization) Events | 32 |
| | 001 | 9.1.5. Statistical Analyses / Methods | |
| | CCI | 004 Fadadat/Wadablaa | 2.4 |
| | | 9.2.1. Endpoint / Variables | |
| | | 9.2.2. Summary Measure | |
| | | 9.2.3. Population of Interest | |
| | | 9.2.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 9.2.5. Statistical Analyses / Methods | 34 |
| 0 | PHAR | MACODYNAMIC ANALYSES | 35 |
| • | 10.1. | Serum Target Engagement Analyses | |
| | | 10.1.1. Endpoint / Variables | |
| | | 10.1.2. Summary Measure | |
| | | 10.1.3. Population of Interest | |
| | | 10.1.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 10.1.5. Statistical Analyses / Methods | 38 |
| | CCI | | |
| | 10.3. | Immunogenicity | 38 |
| | | 10.3.1. Summary Measure | 38 |
| | | 10.3.2. Population of Interest | 39 |
| | (PK/T | MACOKINETIC / TARGET ENGAGEMENT / PHARMACODYNAMIC E/PD) ANALYSES | 39 |
| 2. | | ARKER ANALYSES – PART A ONLY | |
| | 12.1. | Immune Cell Phenotypes | 40 |
| | | 12.1.2. Summary Measure | 40 |
| | | 12.1.3. Population of Interest | 40<br>40 |
| С | CI | 1714 Statistical Analyses / Methods | 41 |
| 13. | REFE | RENCES | 43 |
| | ADDE | NDICEC | 4.5 |
| 14. | | | 45 |
| | 14.1. | 11 | 40 |
| | | Fully Treated Population | 40 |
| | | | AF |
| | 1/1.2 | Protocol Population (Part B) | |
| | 14.2. | •• | |
| | | <b>3</b> | |
| | | 14.2.2. Part A Cohorts With Blister: 0.1 and 0.3 mg/kg IV | |
| | | 14.2.3. Part A Cohorts With Blister: 1 mg/kg IV | |
| | | 14.2.5. Part B | |
| | 1/1/2 | Appendix 3: Assessment Windows | |
| | 14.0. | rippendix o. riaacaament willidowa | |


| -, | п | u | $\mathbf{n}$ |
|----|---|---|--------------|

| 14.4. | Appendix | 4: Study Phases and Treatment Emergent Adverse | |
|---|---|---|---|
| | Events | | .53 |
| | 14.4.1. | Study Phases | .53 |
| | 14.4.2. | Treatment Emergent Flag for Adverse Events | .53 |
| 14.5. | <b>Appendix</b> | 5: Data Display Standards & Handling Conventions | .54 |
| | | Reporting Process | |
| | 14.5.2. | Reporting Standards | . 55 |
| | 1453 | Reporting Standards for Pharmacokinetic | 56 |
| 14.0 | Annondiv | C. Darived and Transformed Data | Ε0 |
| 14.6. | 14.6.1. | 6: Derived and Transformed Data | |
| | 14.6.1. | Study Population | |
| | 14.6.2. | Efficacy | |
| | 14.6.4. | Safety | |
| | | Immunogenicity | |
| 14.7. | | • • | |
| 14.7. | 14.7.1. | 7: Reporting Standards for Missing Data Premature Withdrawals | |
| | 14.7.1. | | |
| 14.0 | | Handling of Missing Data | |
| 14.8. | | 8: Values of Potential Clinical Importance | |
| 14.9. | | PCI Values for Part B | |
| 14.9. | | | . 70 |
| | 14.9.1. | Calculation of SD from Bayesian Repeated Measures model | 70 |
| | 1492 | Model Checking & Diagnostics | |
| 14 11 | | 10: Abbreviations & Trade Marks | |
| | | Abbreviations | |
| | | Trademarks | |
| 14.12 | | 11: List of Data Displays. | |
| | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | | Deliverables | |
| | | Safety Review Table | |
| | | Sample Size Re-estimation table | |
| | | Study Population Tables | |
| | | Safety Tables | |
| | | Pharmacokinetic Tables | 85 |
| | | Pharmacokinetic Figures | |
| | | Pharmacodynamic Tables | |
| | | Pharmacodynamic Figures | |
| | | Biomarker Tables | |
| | | Biomarker Figures | |
| | | Efficacy Tables | |
| | | Efficacy Figures | |
| | | ICH Listings | |
| | | ICH Conditional Listings | |
| | | Non-ICH Listings | |
| | | <b>▽</b> | |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 207804:

| Revision Chronology: | | |
|----------------------|-------------|----------------|
| Amendment 7 | 09-FEB-2022 | TMF-14447953 |
| Amendment 6 | 12-NOV-2021 | TMF-11834237 |
| Amendment 5 | 07-SEP-2020 | 2017N342035_05 |
| Amendment 4 | 14-NOV-2019 | 2017N342035_04 |
| Amendment 3 | 18-JUL-2019 | 2017N342035_03 |
| Amendment 2 | 21-NOV-2018 | 2017N342035_02 |
| Amendment 1 | 10-APR-2018 | 2017N342035_01 |
| Original Protocol | 02-FEB-2018 | 2017N342035_00 |

# 1.1. **Version history**

| SAP<br>Version | Approval<br>Date | Protocol Version<br>(Date) on which<br>SAP is Based | Change | Rationale |
|---|---|---|---|---|
| SAP | 01-MAR-<br>2021 | 2017N342035_05<br>(07-SEP-2020) | Not Applicable | Original version. |
| SAP<br>amendment<br>1 | 01-JUN-<br>2021 | 2017N342035_05<br>(07-SEP-2020) | Part B sections | Part A, unmodified from previous version, and amended Part B. |
| SAP<br>amendment<br>2 | 24-MAR-<br>2022 | TMF-14447953<br>(09-FEB-2022) | Part B Sections Programming notes for PK and TE outputs Adding additional Interim Analyses Information | Protocol was amended to account for two additional Interim Analyses. |
| SAP<br>Amendment<br>3 | 28-JUL-<br>2022 | TMF-14447953<br>(09-FEB-2022) | Primary model update. Clarification on Intercurrent Events section. Additional outputs for IA4 and Part B SAC. Inclusion of safety tables (Part B 2.37-2.39) | Update to the model specification to avoid overparameterization by removal of the random subject intercept, and to include only data during the treatment period (i.e. up to week 8) in the primary analysis model. (Section 7) |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol 2017N342035\_05 [(Dated: 07-Sep-2020)].

# 2.2. Study Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| Parts A and B To evaluate the safety and tolerability of escalating doses of GSK3858279 following single IV, single SC dosing in healthy participants and repeat SC dosing in OA participants. | Adverse Events (AE) and Serious Adverse<br>Events (SAE).<br>Clinical laboratory measurements, 12-lead<br>electrocardiograms (ECG) and vital signs. |
| Part B To assess changes in pain in participants with OA of the knee following repeat SC dosing. | Change from baseline in average knee pain intensity at week 8. Change from baseline in worst knee pain intensity at Week 8. |
| Secondary | |
| To describe the pharmacokinetics (PK) of GSK3858279 following single IV, single SC in healthy participants and repeat SC dosing in OA participants. | CCI |
| To evaluate the target engagement (TE) of CCL17 by GSK3858279 following single IV, single SC dosing in healthy participants and repeat SC dosing in OA participants. | CGI |
| CCI | |



## 2.3. Study Design

This study will be a randomized, double-blind, placebo-controlled, two-part trial. A study diagram is included in Table 1.

Part A will be a single ascending dose escalation study to evaluate the safety, tolerability, PK, and target engagement of GSK3858279 in healthy participants. Single IV doses and a single SC dose will be investigated in separate cohorts of participants. Target engagement will be assessed both in blood and GC

Up to five single ascending IV dose levels of GSK3858279 will be investigated. A single SC dose of GSK3858279 will also be assessed to determine bioavailability, as future studies as well as the target product will likely involve SC administration.

A Dose Escalation Committee (DEC) will review at least 15 days of safety and PK data prior to progression to the next dose level. The decision to progress the SC cohort will be based upon understanding the PK and TE data from some IV cohorts. Once sufficient safety, PK and target engagement data is collected from the top IV dose and SC cohorts, a data review will take place and a decision to proceed with Part B of the study may be made.

In Part A, sentinel participants will be used in each dosing cohort: two participants will be dosed first, one will be randomized to GSK3858279 and one to placebo. 48-hour post dose safety data from the sentinel participants will be reviewed by the investigator and the remainder of the cohort will then be dosed if deemed safe to do so.

Part B will investigate the safety, tolerability, clinical efficacy on pain (as primary endpoints), PK, target engagement and immunogenicity in participants with OA of the knee after weekly SC dosing for 8 weeks of GSK3858279 or placebo in a 1:1 ratio.

The table below provides an overview of the study design and the key features.

#### Table 1 Study Design

#### Study Design

Figure 1: Parts A and B: Study Design



IV: intravenous; N: number of participants; OA: osteoarthritis; PK: pharmacokinetics; SC: subcutaneous

# Part A Design features

- Within each cohort, and hence at each dose level, GSK3858279 and placebo will be administered in a 3:1 ratio according to the randomisation schedule, in a blinded manner.
- Of the eight participants within each cohort, six will receive GSK3858279 and two will receive placebo, as per the randomisation schedule.
- Up to a maximum of 5 IV dose levels and 1 SC dose level will be studied in total in Part A. To mitigate a risk of adverse reactions, sequential dosing will be implemented. Two sentinel participants will receive study intervention first (one on active, one on placebo) per dosing cohort and will be monitored in the clinical unit for approximately 48 hours.
- Assuming adequate safety from these two participants over the first 48 hrs postdose, the remaining participants in the cohort can then be dosed.
- Dose escalation data reviews will occur once sufficient safety and PK data is obtained from a cohort, and a dose escalation to the next planned dose may occur.
- The decision to proceed to the next dose level of GSK3858279 will be made at a Dose Escalation Committee (DEC) meeting. Details are included in the Dose Escalation Plan (DEP).
- Upon review of data from the 1 mg/kg IV cohort, the DEC may decide to trigger the SC cohort as well as the 3 mg/kg IV cohort, if data are satisfactory.
- Once eight participants in the highest dose cohort in Part A have completed the Day 15 visit, the DEC will review all available safety, PK, target engagement (i.e, free and total CCL17 levels) in serum and decide whether to proceed with Part B of the study.

#### Study Design In case of early dropouts, a minimum of 6 participants completing the Day 15 visit will be required for dose escalation data review Based on the emerging PK and TE data from Part A. a single IV dose up to 10 mg/kg is not suitable to test the mechanism in OA participants and hence a repeat SC dose of 240 mg is now considered more appropriate (Protocol Amendment #3. July 2019) and Protocol Amendment #5, Sept 2020 based on the observed TE of 3 mg/kg SC and predicted TE after repeat SC dosing. Part A Time Refer to Appendix 2 & Events Part A Within each cohort, participants will be assigned to either GSK3858279 or placebo in a Treatment 3:1 ratio, where the intervention codes are as follows: sequences Intervention code Intervention Description 0.1 mg/kg IV GSK3858279 0.3 mg/kg IV GSK3858279 В C 1 mg/kg IV GSK3858279 D 3 mg/kg IV GSK3858279 Ε 10 ma/ka IV GSK3858279 F SC GSK3858279 Placebo Part B In Part B, the total duration of the study (from 1st screening visit until final follow-up) Design for each participant will be up to 182 days (inclusive of a screening period of a Features maximum of 42 days). Approximately 50 (up to a maximum of 80) participants with OA will be randomly assigned to GSK3858279 or placebo in a 1:1 ratio. Each participant will receive weekly SC doses of either 240 mg GSK3858279 or placebo for 8 weeks. Close in-stream safety review (AEs, clinical laboratory, vital signs, cardiac monitoring) is planned throughout for all participants (see Safety Management Plan). An early detailed review of safety, PK, TE and ADA data following administration of repeat doses is intended for the first 8 participants (4 randomized to active treatment) when the 8th participant completes the Week 4 assessment. A second detailed review of safety, PK, TE and ADA data is intended for the first 20 participants (10 randomized to active treatment) when the 20th participant completes the Week 4 assessment. An interim analysis for futility will occur once approximately 20 participants have completed the Week 4 assessment. A second interim analysis for an unblinded sample size re-estimation, including a futility assessment, may occur prior to enrolling the 50th participant, where the sample size could be decreased to a minimum of 20 or increased to a maximum of 80 participants enrolled if the observed SD of Change from baseline in the average knee pain intensity at week 8 is smaller or greater than 1.8 respectively. Sample size increase may also occur to account for participants who discontinue the treatment or study prior to Week 8. See Section 7.1.5.1 for more details Additional interim analyses may occur for internal decision making and/or interaction with regulatory agencies as appropriate.

| Study Design | | | |
|---|---|---|---|
| Part B Time | • R | efer to Appendix 2 | |
| & Events | | •• | |
| Part B | • Pa | Participants will be assigned to either GSK3858279 or placebo in a 1:1 ratio, where | |
| Treatment | th | the intervention codes are as follows: | |
| sequences | | | |
| | | Intervention code Intervention Description | |
| | | G 240 mg SC GSK3858279 | |
| | | Р | Placebo |

# 2.4. Statistical Analyses

As the primary objective for part A of the study is safety and tolerability, and for part B is safety, tolerability and efficacy there are no formal hypotheses to be evaluated.

**Part A:** An assessment of dose proportionality will be conducted for selected pharmacokinetic endpoints (*i.e.* Cmax, and  $AUC(0-\infty)$  and/or AUC(0-t)) following single IV dose. In addition, an exploratory comparison will be made between the IV and SC formulations at the dose level studied. This will be only done for the 3 mg/kg IV and SC doses.

**Part B:** A comparison between GSK3858279 and Placebo will be made on the pain numerical rating scale. An assessment will be made comparing GSK3858279 to placebo with respect to the change from baseline in average pain intensity at week 8. The change from baseline in worst pain intensity at week 8 will also be assessed.

#### 3. PLANNED ANALYSES

#### 3.1. **Interim Analyses**

**Part A:** No formal interim statistical analyses are planned. However, dose escalation meetings will occur at a relevant timepoint after each dose level; including between Parts A and B.

The decision to proceed to the next cohort, and next dose strength to be studied, will be made by the Dose Escalation Committee (DEC) based on assessment of safety and serum GSK3858279 pharmacokinetic data obtained in all participants at the prior dose level. Individual safety data (adverse events, laboratory safety tests, ECGs and vital signs) will be reviewed. In addition, immunogenicity data may be reviewed by the DEC during the study. Once sufficient safety, PK and target engagement data is collected from the top IV dose and SC cohorts, a data review will take place and a decision to proceed with Part B of the study may be made. Further details are included in the Dose Escalation Plan (DEP) Version 003 dated 19-Nov-2018.

Unblinded data from Part A may be reported out in full following the last subject last visit in this part of the study and prior to the conclusion of Part B.

**Part B:** The first interim analysis will occur once approximately 20 participants have completed the Week 4 assessment. A second interim analysis for an unblinded sample

size re-estimation may occur prior to enrolling the 50th participant, where the sample size could be decreased to a minimum of 20 or increased to a maximum of 80 participants.

Additional interim analyses may occur in order to inform internal decision making and/or for interaction with regulatory agencies as appropriate.

In addition to the interim analyses, two planned blinded safety data reviews as specified in the protocol will be carried out to decide upon dose adjustment, participant continuation/ discontinuation and if need be, to stop the study due to safety concerns. The necessary unblinded data will be summarised in a blinded fashion either by using dummy participant IDs or by presenting only group level data.

Further details of the part B interim analyses and safety reviews are outlined in the Interim Analysis Charter.

## 3.2. Final Analyses

The final planned analyses (Parts A and B) will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol (Section 4.5 End of Study Definition of the protocol): The end of the study is defined as the date of the last visit (including follow-up) of the last participant in the study (Parts A and B).
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management. The final delivery for Part A may be generated in its own reporting area prior to the completion of Part B of the study once Data Management has declared DBF for Part A. Parts A and B final deliveries may be generated and kept in separated reporting areas.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG and RAMOS NG procedures.

# 4. ANALYSIS POPULATIONS

# 4.1. **Analysis Populations**

# 4.1.1. Part A and B

| Population | Description | Outputs |
|---|---|---|
| Screened | All participants who were screened for eligibility | Study Population<br>(specific only) |
| Enrolled | All participants who passed screening and entered the study. | Study Population<br>(Specific only) |
| | <ul> <li>Note screening failures (who never passed<br/>screening even if rescreened) and participants<br/>screened but never enrolled into the study are<br/>excluded from the Enrolled population as they did<br/>not enter the study.</li> </ul> | |
| Randomized | <ul> <li>All participants who were randomly assigned to treatment in the study.</li> <li>This population will be based on the treatment the participant was randomized to.</li> </ul> | Study Population |
| Safety | <ul> <li>All randomized participants who received at least one dose of study treatment.</li> <li>This population will be based on the treatment the participant received.</li> </ul> | <ul><li>Study Population<br/>(specific only)</li><li>Safety</li><li>PD</li></ul> |
| Pharmacokinetic | <ul> <li>All participants in the Safety population who had at least 1 reportable serum PK assessment.</li> <li>This population will be based on the treatment the participant received.</li> <li>Note: Non-quantifiable [NQ] values will be considered as reportable values</li> </ul> | • PK |

# 4.1.2. Part A only

| Population | Description | Outputs |
|---|---|---|
| Blister | <ul> <li>All participants in the Safety population who had at least one blister assessment.</li> <li>This population will be based on the treatment the participant received.</li> </ul> | • PD |
| Blister<br>Pharmacokinetic | <ul> <li>All participants in the Safety population who had at least 1 reportable blister PK assessment.</li> <li>This population will be based on the treatment the participant received.</li> </ul> | • PK |

| | Note: Non-quantifiable [NQ] values will be | |
|---|---|---|
| cci | | |
| Fully treated | <ul> <li>All participants in the Safety population who<br/>received at least 80% of planned study<br/>treatment*.</li> </ul> | PK, PD |
| | <ul> <li>This population will be identified by review of<br/>protocol deviations</li> </ul> | |

<sup>\*</sup>Part A has a single dose. Percentage of actual amount administered will be derived using the planned dose and the injected infusion volume.

#### 4.1.3. Part B only

| Population | Description | Outputs |
|---|---|---|
| Intent-to-Treat | <ul> <li>All randomized participants who received at least one dose of study treatment.</li> <li>This population will be based on the treatment the participant was randomized to. Any participants who receive a treatment randomization number will be considered to have been randomized. </li> </ul> | Efficacy |
| Per Protocol | <ul> <li>All participants in the ITT population who comply with the protocol.</li> <li>Protocol deviations that would exclude participants from the PP population are defined in Section 4.2 (Protocol Deviations) and Appendix 1: Exclusions from Per Protocol Population*).</li> </ul> | Efficacy<br>(specific only) |

<sup>\*</sup> This population will be based on the treatment the participant was randomized to.

#### 4.2. Protocol Deviations

Important protocol deviations (including but not limited to deviations related to study inclusion/exclusion criteria, and additionally in part B: prohibited medications, rescue medications, study medication and missing diary data) will be summarised and listed.

Important deviations which result in exclusion from the analysis population will also be summarised and listed.

Please refer to Appendix 1.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

 Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.


207804

• This dataset will be the basis for the listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This output will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

#### 5.1. **General**

Separate outputs will be generated for both Part A and Part B.

## 5.2. Study Treatment Display Descriptors

In the Tables, Listings and Figures (TLF), treatment should be presented with placebo first, then in order of increasing dose by route of administration within each part.

| Part A: Treatment group descriptions | | | |
|---|---|---|---|
| RandAll NG | | Data displays for reporting | |
| Code Description | | Description | Order in TLF |
| Α | 0.1 mg/kg IV GSK3858279 | 0.1 mg/kg IV GSK3858279 | 2 |
| В | 0.3 mg/kg IV GSK3858279 | 0.3 mg/kg IV GSK3858279 | 3 |
| С | 1 mg/kg IV GSK3858279 | 1 mg/kg IV GSK3858279 | 4 |
| D | 3 mg/kg IV GSK3858279 | 3 mg/kg IV GSK3858279 | 5 |
| Е | 10 mg/kg IV GSK3858279 | 10 mg/kg IV GSK3858279 | 6 |
| F | SC GSK3858279 | 3 mg/kg SC GSK3858279 | 7 |
| Р | Placebo | Placebo | 1 |

| Part B: Treatment group descriptions | | | |
|---|---|---|---|
| RandAll | RandAll NG Data displays for reporting | | |
| Code Description | | Description | Order in TLF |
| G | 240 mg SC GSK3858279 | 240 mg SC GSK3858279 | 2 |
| Р | Placebo | Placebo | 1 |

#### 5.3. Baseline Definitions

The baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline. Replicate assessments at a timepoint will be averaged, and the mean value will be used. Unless otherwise stated, if baseline data is missing, no derivation will be performed and baseline will be set to missing.

For the average and worst knee pain intensity, the mean of the scores in index knee over 7 days prior to dosing (Day -7 to Day -1) will be considered as baseline. Baseline should be calculated only if pain scores are recorded on at least 5 days out of 7. If pain scores are not recorded on at least 5 days, the baseline will be set to missing.

For Part B of the study, the CCL17 levels (free, total) baseline value will be derived by averaging the two pre-dose measurements (i.e., average of Day-4 and Day 1).

# 5.4. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices

| Section | Component |
|---|---|
| Section 14.3 | Appendix 3: Assessment Windows |
| Section 14.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| Section 14.5 | Appendix 5: Data Display Standards & Handling Conventions |
| Section 14.6 | Appendix 6: Derived and Transformed Data |
| Section 14.7 | Appendix 7: Reporting Standards for Missing Data |
| Section 14.8 | Appendix 8: Values of Potential Clinical Importance |

# 6. STUDY POPULATION ANALYSES

The study population analyses will be based on the Randomized population, unless otherwise specified.

Study population analyses including analyses of participants' disposition, protocol deviations, demographic characteristics, prior and concomitant medications, baseline efficacy parameters, exposure, medical history and substance use will be based on GSK Core Data Standards.

Details of the planned displays are presented in Appendix 11.

#### 7. EFFICACY ANALYSES – PART B ONLY

# 7.1. Co-primary Efficacy Analyses

## 7.1.1. Endpoint / Variables

The changes in pain in participants with OA of the knee following repeat SC administration are assessed using:

- Change from baseline in the average knee pain intensity at week 8.
- Change from baseline in the worst knee pain intensity at week 8.

# 7.1.2. Summary Measure

The primary summary measure will be the difference between treatments in mean change from baseline. The pain scores will be listed by participant and summarized descriptively by treatment.

#### 7.1.3. Population of Interest

The analyses will be based on the Intent-to-Treat population, unless otherwise specified.

# 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

There is one intercurrent event that is of interest:

1. Treatment Withdrawal (Participant discontinues the study treatment but continues to stay in the study)

No imputations would be carried out if there are missing data due to intercurrent events.

A hypothetical strategy will be used to estimate what the treatment effect would have been had the subject not experienced the intercurrent event. Data collected after the occurrence of the Intercurrent Event will be listed but not used in summary stats and stats analysis TFLs. Since the dosing interval in this study is 7 days, the date of occurrence of the treatment withdrawal intercurrent event will be defined as the date of the first missed dose of study treatment i.e. date of last dose of study treatment + 7 days. Pain scores are measured daily in the evening, therefore pain scores on or after the date of last dose of study treatment + 7 days will be considered as occurring after treatment withdrawal.

#### 7.1.5. Statistical Analyses / Methods

#### 7.1.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

- Change from baseline in Average Knee Pain Intensity at Week 8
- Change from baseline in Worst Knee Pain Intensity at Week 8

## **Model Specification**

- A Bayesian repeated measures model will be used to fit the change from baseline from Week 1 to Week 8.
- The endpoints will be assumed to follow a multivariate (MVN) normal distribution to model all repeated measurements within the same participant.
- Markov-Chain-Monte-Carlo (MCMC) method will be used to estimate the posterior distributions.
- A linear model for Change from Baseline at each Week (visit) will be constructed to model the within-participant covariance structures.
- Terms fitted in the model will include:
  - Categorical: Week (Week 1 to Week 8), Treatment (GSK3858279 and placebo), Treatment\*Week Interaction, Baseline\*Week Interaction
  - Continuous: Baseline
  - o Repeated: Week
- The prior for the Variance Covariance Matrix will follow an Inverse Wishart Distribution.
- Vague priors (normal (0, var=1e6)) will be used for all other model parameters.
- Set simulation size at a minimum of 10000 and 1000 burn-in iterations. The simulation size and number of burn-in iterations could be updated during the convergence check.
- Refer to Appendix 6 Bayesian Repeated Measures Model (PROC MCMC) for additional information
- Refer to Appendix 3 for details on visit computation.
- Refer to Appendix 9 for additional information

## **Model Checking & Diagnostics**

- Bayesian Analyses: Refer to the relevant documentation (Bayesian Statistics Best Practice at GSK – Clinical Trials using Bayesian Inference).
- Refer to Appendix 9

#### Model Results Presentation

- Medians and 95% credible intervals will be produced by treatment group and for the difference between treatment groups, for each of the endpoints,
- The posterior distributions will be used to produce several probability statements:
  - P[True Difference (GSK3858279 placebo) < X</li>
  - o where values of X to be generated are 0, -0.6, -0.8 and -1.0
- For all tables/figures presenting results from a statistical model, a footnote including model, prior distributions, covariates and a very brief mention of intercurrent events will be added.
- For all TFLs presenting efficacy endpoints, a footnote to state a range of the score for the endpoint specifying which direction of change is an improvement.

#### **Interim Analysis 1**

- A first interim analysis will occur once 20 participants reach Week 4
- The endpoint will be Change from baseline in average knee pain intensity at week 4

#### **Interim Analysis 2**

- A second interim analysis may occur once approximately 45 participants have been randomised (this estimated to happen when 28 participants reach Week 8) and will include a sample size re-estimation and a futility assessment. In addition to posterior probabilities, predictive probabilities of achieving criteria of interest at the end of the study will be estimated using a Bayesian Normal-Normal update. Vague priors for all modelling parameters will be used to compute the posterior distributions.
- Criteria of interest are:
  - P[True Difference (GSK3858279 placebo) < X] where values of X to be generated are 0, -0.6, -0.8 and -1.0 and
  - Predictive probability > X%
- At the interim analysis an estimate of the standard deviation of the endpoint at week 8
  will be estimated from the Bayesian Repeated Measures model. Details are given in
  Section 14.9.1. All data available at the time of the interim will be used for this purpose
- The ratio of the Estimated SD to Predicted SD (SD=1.8) for the change from baseline at Week 8 will be used to calculate the optimal sample size as follows:

$$SS_{optimal} = \left(\frac{SD_{estimated}}{1.8} \times \sqrt{50}\right)^2$$

The optimal sample size must be within the range [# participants randomised, 80] subjects (i.e. if the optimal calculation is >80, the SS will be capped at 80/ if the optimal calculation is <50, the SS will be capped at # participants randomised). The number of participants resulting from the SS\_optimal formula must be rounded up to the next even number.</li>

#### Subgroup Analyses

No subgroup analysis is planned for the study.

#### **Sensitivity Analyses**

Refer to Section 14.9.2 for additional information.

#### **Supportive Analyses**

The Bayesian Repeated Measures Model will be performed on the Per Protocol Population if the Per Protocol Population comprises 50 to 90% of the ITT population



## 7.2.2. Summary Measure

The difference in treatment mean change from baseline for WOMAC subscales scores and will be analysed. In addition, the absolute and change from baseline values of WOMAC subscales scores, and colored (Individual and Overall) will be summarized descriptively by treatment. These scores will be also be listed by each participant and treatment.

Refer to Section 14.6.3 for details on calculation of WOMAC subscales scores.

The number of participants who took rescue medication will be summarised by treatment. In addition, the total weekly dose, average weekly dose and average rescue medication use will be summarized. A listing of rescue medication will be produced.

#### 7.2.3. Population of Interest

The efficacy analyses will be based on the Intent-to-Treat population, unless otherwise specified.

#### 7.2.4. Strategy for Intercurrent (Post-Randomization) Events

#### Intercurrent Events:

 Treatment Withdrawal (Participant discontinues the study treatment but continues to stay in the study)

No imputations will be carried out if there are missing data due to intercurrent events.

A hypothetical strategy will be used to estimate what the treatment effect would have been had the subject not experienced the intercurrent event. Data collected after the occurrence of the Intercurrent Event will therefore not be used in the analysis. Since the dosing interval in this study is 7 days, the date of occurrence of the treatment withdrawal intercurrent event will be defined as the date of the first missed dose of study treatment

i.e. date of last dose of study treatment + 7 days. WOMAC, and PainDetect are measured pre-dose at each weekly visit, therefore assessments after the date of last dose of study treatment + 7 days will be considered as occurring after treatment withdrawal. Rescue Medication is assessed daily in the evening, therefore Rescue Medication on or after the date of last dose of study treatment + 7 days will be considered as occurring after treatment withdrawal.

#### 7.2.5. Statistical Analyses / Methods

#### 7.2.5.1. Statistical Methodology Specification

#### Endpoint / Variables

WOMAC pain, stiffness and function subscales scores at Week 1,2,4,6,8

## Model Specification

- A Bayesian repeated measures model will be used to fit the change from baseline from Week 1 to Week 8.
- The endpoints will be assumed to follow a multivariate (MVN) normal distribution to model all
  repeated measurements within the same participant.
- Markov-Chain-Monte-Carlo (MCMC) method in SAS will be used to estimate the posterior distributions of the endpoints.
- A linear model for Change from Baseline at each Week (visit) will be constructed to model the within-subject covariance structures.
- Terms fitted in the model will include:
  - Categorical: Week, Treatment (GSK3858279 and placebo), Treatment\*Week Interaction, Baseline\*Week Interaction
  - Continuous: Baseline
  - Repeated: Week
- The prior for the Variance Covariance Matrix will follow an Inverse Wishart Distribution.
- Set simulation size at a minimum of 10000 and 1000 burn-in iterations. The simulation size and number of burn-in iterations could be updated during the convergence check.
- The vague priors (normal (0, var=1e6)) will be used for the hyperparameters/all model parameters
- •
- Refer to Appendix 6 Bayesian Repeated Measures Model (PROC MCMC) for additional information
- Refer to Appendix 3 for details on visit computation.
- Refer to Appendix 9 for additional information

#### Model Checking & Diagnostics

- Bayesian Analyses: Refer to the relevant documentation (Bayesian Statistics Best Practice at GSK – Clinical Trials using Bayesian Inference).
- Refer to Appendix 9

#### Model Results Presentation

 Medians and 95% credible intervals will be produced by treatment group and for the difference between treatment groups each of the endpoints

- The posterior distributions will be used to produce several probability statements:
- For WOMAC pain, stiffness and function subscales scores
  - P[True Difference (GSK3858279 placebo) < X] where values of X to be generated are 0, -0.6, -0.8 and -1.0



 For all tables/figures presenting results from a statistical model, a footnote including model, prior distributions, covariates and a very brief mention of intercurrent events will be added.

 For all TFLs presenting efficacy endpoints, a footnote to state a range of the score for the endpoint specifying which direction of change is an improvement.

#### Subgroup Analyses

No subgroup analyses is planned for the study.

#### SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

# 8.1. Adverse Events Analyses

The definition of an AE is detailed in Appendix 3 of the protocol (Section 10.3).

Analyses of AEs will include those events that are on-treatment (Section 14.4.1).

Adverse events analyses including the analysis of Adverse Events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards.

Details of the planned displays are presented in Appendix 11.

# 8.2. Clinical Laboratory Analyses

Laboratory evaluations will be based on GSK Core Data Standards and will include:

- Hematology laboratory tests
- Chemistry laboratory tests
- Urinalysis
- Other screening tests

Details of the planned displays are presented in Appendix 11.

The laboratory assessments for each category are displayed in Table 2.

 Table 2
 Laboratory Assessments

| Laboratory<br>Assessments | Parameters | | | | | |
|---|---|---|---|---|---|---|
| Hematology | Platelet Count | | RF | BC Indices: | WBC count with Differential: | |
| Tiomatology | RBC Count | | MC | | Neutrophils | |
| | Hemoglobin | | | CH | Lymphocyte | • |
| | Hematocrit | | %Reticulocytes | | Monocytes | |
| | ricinatocht | | | | Eosinophils | |
| | | | | | Basophils | |
| Clinical | BUN | Potassiu | m | Aspartate Amino | | Total and direct |
| Chemistry <sup>1,2,3</sup> | | | | (AST)/ Serum GI | utamic- | bilirubin |
| | | | | Oxaloacetic Trar | nsaminase | |
| | | | | (SGOT) | | |
| | Creatinine | Sodium | | Alanine Aminotransferase | | Total Protein |
| | | | | (ALT)/ Serum Gl | | |
| | | | | Pyruvic Transaminase | | |
| | | 0.1. | | (SGPT) | | 20 1: |
| | Glucose (non-fasting) Calcium | | | Alkaline phospha | atase | <sup>2</sup> Cardiac |
| | | | | | | troponin T |
| Routine | Specific gravity | , | | | | <sup>3</sup> NT-proBNP |
| Urinalysis <sup>1</sup> | | · | nd l | retones hiliruhin i | ırohilinoden | nitrite leukocyte |
| Officialysis | pH, glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase by dipstick | | | | | |
| | Microscopic examination and laboratory quantification of proteinuria (if | | | | | |
| blood or protein is abnormal on dipstick) | | | | | ( | |
| | Part B: Alcohol | | | | | |
| Combined | 7 (1) 2.7 (30)(0) | | | | | |
| throat and | COVID-19 (SARS-CoV2) (see SRM for further details) | | | | | |
| nasopharyngeal | , , , | | | | | |
| swab | | | | | | |
| Other | Blood (serum): | | | | | |
| Screening | | • | | and estradiol (as r | needed in wo | men of non- |
| Tests childbearing potential only) Serology (TB test, HIV antibody, HBsAg, HBcAb and hepatitis C vi | | | | | | |
| | | | | | tis C virus | |
| | antibody) | | | | | |
| | QuantiFERON test | | | | | |
| | Complement protein C3 and C4 Urine: Urine drug screen to include at minimum: amphetamines, barbiturates, | | | | | |
| | | | | | | arhiturates |
| | _ | | | ds and benzodiaze | | arbituratos, |
| | Urine albumin- | | | | 7pii 100. | |

#### Notes

1. Details of liver chemistry stopping criteria and required actions and follow-up assessments after liver stopping or monitoring event are given in Protocol Section 7.2.1 and Appendix 6a and 6b of protocol. All events of ALT  $\geq$ 3 × upper limit of normal (ULN) and bilirubin  $\geq$ 2 × ULN (>35% direct bilirubin) or ALT  $\geq$ 3 × ULN and international normalized ratio (INR) >1.5, if INR measured, which


207804

may indicate severe liver injury (possible Hy's Law), must be reported as an SAE (excluding studies of hepatic impairment or cirrhosis).

- 2. Troponin T using high sensitivity test.
- 3.NT-proBNP (N-terminal pro B-type natriuretic peptide) at baseline and Day 57 visit only.

Laboratory/analyte results that could unblind the study will not be reported to investigative sites or other blinded personnel until the study has been unblinded.

## 8.3. Other Safety Analyses

The analyses of non-laboratory safety test results will be based on GSK Core Data Standards, unless otherwise specified.

The non-laboratory safety test results include:

- Vital Signs
- ECGs
- Echocardiogram
- Telemetry (for Part A only)
- Holter monitoring (for Part B only at Screening)

# 8.4. **COVID-19 Pandemic Statistical Displays**

A summary of the following COVID-19 assessments may be produced: Case Diagnosis, COVID-19, Test performed, and Results of the COVID-19 test. Additionally, a listing of all subjects with visits and assessments impacted by the pandemic may be produced. The listing will include:

- 1. Site Identifier
- 2. Treatment for parallel group studies
- 3. Unique Subject Identifier
- 4. Subject Identifier
- 5. Impacted Visit
- 6. Impact
- 7. Reason for Impact

Details of the planned displays are presented in Appendix 11.

# 9. PHARMACOKINETIC ANALYSES

#### 9.1. Serum Pharmacokinetics

The PK analyses described below will be carried out for GSK3858279 in serum.

# 9.1.1. Endpoint / Variables

CCI

# 9.1.1.1. Drug Concentration Measures

Refer to Appendix 5(Section 14.5.3).

#### 9.1.1.2. Derived Pharmacokinetic Parameters



NOTES:



#### 9.1.1.2.2. Part B



Additional parameters may be included as required.

In the event that a robust and predictive population PK/TE model cannot be developed e.g. data limited by high levels of NR data, all parameters listed in the table will be derived directly from the observed data using standard non-compartmental analysis. In such case, PK parameters for subjects on sparse sampling schedule will be only calculated at weeks 1 and 8.

# 9.1.2. Summary Measure

Individual and mean/median concentration-time profiles of GSK3858279 in serum (stratified by treatment group in Part A) will be plotted and listed. Serum concentrations will be summarized descriptively. Derived serum PK parameters will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 9.1.3. Population of Interest

The serum pharmacokinetic analyses will be based on the Pharmacokinetic population, unless otherwise specified.

## 9.1.4. Strategy for Intercurrent (Post-Randomization) Events

Missing data would be considered as Missing at Random and no imputations for missing data would be carried out.

## 9.1.5. Statistical Analyses / Methods

Details of the planned displays are presented in Appendix 11 and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 9.1.5.1. Dose proportionality

Dose proportionality in Part A will be assessed by visual inspection of:

 Dose normalised AUC(0-∞) [or if not available AUC(0-t)] and Cmax values versus dose.

Dose proportionality may also be assessed using the power model described below.

#### Dose proportionality

#### **Endpoints**

• AUC(0-t), AUC(0-∞) and Cmax

## **Model specification**

Power model (log-log linear model):

$$y = \alpha \times dose^{\beta} \iff \log_e(y) = \log_e(\alpha) + \beta \times \log_e(dose)$$

Where

- o y = endpoint of interest
- o dose = actual dose (mg) received under fasted condition
- β = parameter associated to dose (slope)

- α = subject-specific random effect (intercept)
- Terms fitted in the power model:
  - Response: log transformation of the endpoint of interest log<sub>e</sub>(y)
  - Fixed continuous covariates: log<sub>e</sub>(dose)
  - Random: subject

#### Model checking & diagnostics

- Normality assumptions underlying the model used for analysis will be examined by obtaining a
  normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e.
  checking the normality assumption and constant variance assumption of the model,
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data

# Model results presentation

Table of the estimated slopes and 90% CI (slope close to 1 implies dose proportionality)





#### 9.2.1. Endpoint / Variables

Blister concentrations of GSK3858279.

#### 9.2.1.1. Drug Concentration Measures

Refer to Appendix 5 (Section 14.5.3).

#### 9.2.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will not be calculated due to the sparsity of blister fluid samples.

The within subject and timepoint blister fluid:serum concentration ratio for GSK3858279 may be determined from the concentration-time data if data permit.

#### 9.2.2. Summary Measure

Individual and mean/median concentration-time profiles of GSK3858279 in blister fluid (stratified by treatment group) will be plotted and listed. Blister fluid concentrations will be summarized descriptively.

#### 9.2.3. Population of Interest

The blister pharmacokinetic analyses will be based on the Blister Pharmacokinetic population, unless otherwise specified.

#### 9.2.4. Strategy for Intercurrent (Post-Randomization) Events

Missing data would be considered as Missing at Random and no imputations for missing data would be carried out.

#### 9.2.5. Statistical Analyses / Methods

Details of the planned displays are presented in Appendix 11 and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed

# 10. PHARMACODYNAMIC ANALYSES

#### 10.1. Serum Target Engagement Analyses

The Target Engagement analyses described below will be carried out for Free and Total CCL17 in Serum.

## 10.1.1. Endpoint / Variables

Free and Total CCL17 levels in serum and derived Target Engagement parameters.

#### 10.1.1.1. Target Engagement Concentration Measures

Refer to Appendix 5 (Section 14.5.4).

#### 10.1.1.2. Derived Target Engagement Parameters

#### 10.1.1.2.1. Part A

All Target Engagement parameters in Part A will be determined directly from the observed concentration-time data, as data permits. All calculations will be based on actual sampling times.

Target Engagement parameters that will be calculated for free CCL17 in Part A are listed below. Additional parameters may be included as required.



#### NOTES:

Additional parameters may be included as required.
Target engagement parameters that will be calculated for total CCL17 in Part A are listed below. Additional parameters may be included as required.



NOTES:

Additional parameters may be included as required.

#### 10.1.1.2.2. Part B

All Target Engagement parameters in Part B will be calculated using a model based posthoc analysis and the currently supported version of NONMEM. The model based posthoc analysis is described in Section 11. All calculations will be based on actual sampling times.

Target Engagement parameters that will be calculated for free CCL17 in Part B are listed






#### NOTES:

Additional parameters may be included as required.

<sup>1</sup>In the event that a robust and predictive population PK/TE model cannot be developed e.g. data limited by high levels of NR data, TE parameters will be derived directly from the observed data.

Target engagement parameters that will be calculated for total CCL17 in Part B are listed below. Additional parameters may be included as required.



NOTES:

Additional parameters may be included as required.

<sup>1</sup>In the event that a robust and predictive population PK/TE model cannot be developed e.g. data limited by high levels of NR data, TE parameters will be derived directly from the observed data.

#### 10.1.2. Summary Measure

Individual and median/mean concentration-time profiles of Free and Total CCL17 (stratified by treatment group in Part A) will be plotted and listed. Free and Total CCL17 concentrations in serum will be summarized descriptively.

Derived serum TE parameters will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 10.1.3. Population of Interest

The target engagement analyses will be based on the Safety population, unless otherwise specified.

#### 10.1.4. Strategy for Intercurrent (Post-Randomization) Events

Missing data will not be imputed, regardless the reasons.

#### 10.1.5. Statistical Analyses / Methods

Details of the planned displays are presented in Appendix 11 and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 10.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.



The within subject and timepoint blister fluid:serum concentration ratio for free and total CCL17 may be determined from the concentration-time data if data permit. The free and total CCL17 concentrations will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 10.3. Immunogenicity

#### 10.3.1. Summary Measure

The number and percentage of confirmed positive samples in each treatment group will be presented at each time assessed. Only binding antibody detection is collected in this study. Neutralising antibody detection is not collected.

#### 10.3.2. Population of Interest

The immunogenicity analyses will be based on the safety population, unless otherwise specified.

For the in-stream safety reviews 1 and 2, subject data will be anonymised as outlined in Appendix 6

# 11. PHARMACOKINETIC / TARGET ENGAGEMENT / PHARMACODYNAMIC (PK/TE/PD) ANALYSES

The primary goal of this analysis is to characterize the Pharmacokinetic / Target Engagement (PK/TE) relationship of GSK3858279 following IV and SC administration to healthy and OA participants. The influence of subject demographics and baseline characteristics, including disease activity, may be investigated. PK and TE data will be analysed using the currently supported version of NONMEM. Details of this analysis are described in a separate RAP [GSK Document number TMF-14343601.

The relationship between Pharmacokinetic / Target Engagement / Pharmacodynamic (PK/TE/PD) of GSK3858279 following repeat SC administration to OA participants may also be explored. Details of this analysis are described in a separate RAP GSK Document number TMF-14343601.

# 11.1. Pharmacokinetic / Target Engagement / Pharmacodynamic Dataset Specification

The dataset specification to support any PK/TE/PD analysis will be provided as a separate document.

The merging of PK, TE, treatment, demographic and efficacy data together with the creation of the NONMEM-specific dataset will be performed by, or under the direct auspices of, Clinical Statistics & Programming, GSK.

This dataset programming will be conducted in a HARP environment using the currently supported version of SAS.

#### BIOMARKER ANALYSES – PART A ONLY

#### 12.1. Immune Cell Phenotypes



#### 12.1.2. Summary Measure

Two summary measures are of interest, the treatment effect (Placebo vs GSK3858279) and the difference between sample types (Blood vs Blister).

- Mean Treatment Difference in Change from baseline at all visits
- The within subject and timepoint ratio of Blister:Blood at all visits only for blister induced cohorts of Part A

Measures of sample reliability (Blister Volume and Total White Blood Cell Count) will be listed only.



#### 12.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11 and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 10.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 12.1.4.1. Statistical Methodology Specification

#### **Endpoint / Variables**

Percentage of Immune Cell Phenotypes

#### **Model Specification**

- Endpoints will be analyzed for each flow cytometry cell type using generalized linear mixed models (GLMM) with appropriate link functions or transformations performed as required.
- Terms in GLMM model will include:
  - categorical: baseline, treatment group, sample type, visit and two 3-way interactions
    - baseline with sample type with treatment group
    - visit with sample type with treatment group
  - Random effect: subject
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the RANDOM line.
  - In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.
  - Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- LS Means for the Sample Type by Treatment by Visit will be calculated using the observed baseline mean for each sample type separately.

#### Model Checking & Diagnostics

- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

#### Model Results Presentation

For summary measure 1 (mean treatment difference), for each sample type and each treatment group:

- Number of subjects in analyses
- Least Squares Mean of Change from Baseline with Standard Error

For all GSK3858279 arms

- Difference to Placebo, 95% Confidence Interval and p-value
- In addition for 3 mg SC:
- Difference to 3mg IV, 95% Confidence Interval.

For summary measure 2 (Mean Sample Type Difference), for each treatment group and overall (see note) and each sample type:

- Number of subjects in analyses
- Least Squares Mean of Change from Baseline with Standard Error

For Blister

Difference to Blood, 95% Confidence Interval

Note: overall (treatment-independent) mean will be calculated for Blister and Blood, for each visit.

Plots of LS Means (+/- SE) and Difference (95% CI) will be presented.

## Sensitivity and Supportive Analyses

• A characterisation of the dose and/or exposure response may be carried out if data allows.



#### 13. REFERENCES

GlaxoSmithKline Document Number 2017N342035\_00. Study ID 207804: A two-part phase I randomized double blind (sponsor open) placebo controlled study to evaluate safety, tolerability, pharmacokinetics, target engagement and potential for efficacy of single intravenous and subcutaneous doses of GSK3858279 in healthy volunteers and participants with osteoarthritis of the knee.

GlaxoSmithKline Document Number 2017N342035\_01. Study ID 207804: A two-part phase I randomized double blind (sponsor open) placebo controlled study to evaluate safety, tolerability, pharmacokinetics, target engagement and potential for efficacy of single intravenous and subcutaneous doses of GSK3858279 in healthy volunteers and participants with osteoarthritis of the knee.

GlaxoSmithKline Document Number 2017N342035\_02. Study ID 207804: A two-part phase I randomized double blind (sponsor open) placebo controlled study to evaluate safety, tolerability, pharmacokinetics, target engagement and potential for efficacy of single intravenous and subcutaneous doses of GSK3858279 in healthy volunteers and participants with osteoarthritis of the knee.

GlaxoSmithKline Document Number 2017N342035\_03. Study ID 207804: A two-part phase I randomized, double blind, placebo controlled study to evaluate safety, tolerability, pharmacokinetics and target engagement of single intravenous and subcutaneous doses of GSK3858279 in healthy participants and to evaluate the efficacy of repeat subcutaneous doses in participants with osteoarthritis of the knee.

GlaxoSmithKline Document Number 2017N342035\_04. Study ID 207804: A two-part phase I randomized, double blind, placebo controlled study to evaluate safety, tolerability, pharmacokinetics and target engagement of single intravenous and subcutaneous doses of GSK3858279 in healthy participants and to evaluate the efficacy of repeat subcutaneous doses in participants with osteoarthritis of the knee.

GlaxoSmithKline Document Number 2017N342035\_05. Study ID 207804: A two-part phase I randomized, double blind, placebo controlled study to evaluate safety, tolerability, pharmacokinetics and target engagement of single intravenous and subcutaneous doses of GSK3858279 in healthy participants and to evaluate the efficacy of repeat subcutaneous doses in participants with osteoarthritis of the knee.

GlaxoSmithKline Document Number TMF-11834237. Study ID 207804: A two-part phase I randomized, double blind, placebo controlled study to evaluate safety, tolerability, pharmacokinetics and target engagement of single intravenous and subcutaneous doses of GSK3858279 in healthy participants and to evaluate the efficacy of repeat subcutaneous doses in participants with osteoarthritis of the knee.

GlaxoSmithKline Document Number TMF- 14447953. Study ID 207804: A two-part phase I randomized, double blind, placebo controlled study to evaluate safety, tolerability, pharmacokinetics and target engagement of single intravenous and subcutaneous doses of GSK3858279 in healthy participants and to evaluate the efficacy of repeat subcutaneous doses in participants with osteoarthritis of the knee.


207804

GlaxoSmithKline Document Number TMF-14343601 (v1.0). Project Data Analysis Plan for an Integrated Analysis of GSK3858279 Pharmacokinetic/Target Engagement/Pharmacodynamic relationship in Healthy Participants, Participants with Osteoarthritis of the Knee and other Indications. Effective Date 30-Dec-2021.

#### 14. APPENDICES

# 14.1. Appendix 1: Protocol Deviation Management and Definitions for Fully Treated Population

# 14.1.1. Exclusions from Fully Treated Population (Part A) and Per Protocol Population (Part B)

Part A: A participant meeting any of the following criteria will be excluded from the Fully Treated population:

| Exclusion Description |
|------------------------------------------------------|
| Patient did not receive ≥ 80% of planned medication* |

<sup>\*</sup>Part A has a single dose. Percentage of actual amount administered will be derived using the planned dose and the injected infusion volume. In case a subject didn't receive a full dose in PART A, the actual amount of drug administered (AMT) will be calculated as AMT [mg]= numerical part of treatment group [mg/kg] \* WTBL [kg] \* percentage of infusion volume / 100 when EXPOSURE.ACTTRT is "GSK3858279". In case a subject from the 3 mg/kg SC treatment group didn't receive a full dose and WTBL≥ 80 kg, then AMT [mg]= 240 [mg] \* percentage of infusion volume / 100. The percentage of infusion volume (TVOLPCT) is assumed 100 for a full dose.

Part B: A participant who meets any of the below criteria will be excluded from the Per Protocol population:

| Violation<br>Category | Criterion<br>Violated | Deviation |
|---|---|---|
| Inclusion/<br>Exclusion<br>Criteria | Inclusion Criteria<br>No. 7 | Did not have OA of the index knee as defined by symptoms for ≥6 months with a clinical diagnosis of OA as per American College of Rheumatology (ACR) clinical diagnosis criteria |
| | Inclusion Criteria<br>No. 8 | Did not have an average of daily pain score ≥4 and ≤9 by the 11-point NRS (0-10) in index knee over 7 days prior to dosing (Day-7 to Day-1). Data should be recorded on at least 5 of 7 occasions by the participant to obtain a valid baseline value. |
| | Inclusion Criteria<br>No. 9 | Did not have a Kellgren and Lawrence (KL) score ≥2 on X-ray obtained during screening (Kellgren, 1957). |
| | Exclusion<br>Criteria No. 39 | Diagnosis of current inflammatory arthritis such as rheumatoid arthritis, autoimmune disorder affecting joints, seronegative spondyloarthritis, gout or pseudogout in any joint (defined as acute episodic attacks of swollen, painful joint in a patient with X-Ray chondrocalcinosis or calcium pyrophosphate dihydrate [CPPD] crystals). Note: asymptomatic CPPD crystals on X-ray are not an exclusion |
| | Exclusion<br>Criteria No. 67 | Underwent intra-articular therapy within 3 months prior to signing the informed consent. |
| | Exclusion<br>Criteria No. 68 | Intake of Immunosuppressants, including corticosteroids (parenteral within 3 months of screening; oral within 1 month of screening). |
| Prohibited<br>Medications* | | Any use of Systemic Corticosteriods from screening until the end of Week 8 |

| Violation | Criterion | Deviation |
|---|---|---|
| Category | Violated | Any use of Intro-orticular thorapy of the index joint from |
| | | Any use of Intra-articular therapy of the index joint from |
| | | screening until the end of Week 8 |
| | | Any use of, opioids, NSAIDs, topical analgesics or anti- |
| | | neuropathic agents 24 hours before a clinical visit on more |
| | | than 1 visit during the first 8 weeks (Day 1 – Day 57) |
| | | Any use of opioids, NSAIDs, topical analgesics or anti- |
| | | neuropathic agents for more than 1 day per week on more |
| | | than 1 visit during the first 8 weeks (Day 1 – Day 57) |
| CCI | | |
| Study | | Missing more than 1 dose out of 8 doses of study treatment |
| Medication | | |
| Missing | | Missing average knee pain or worst knee pain diary data for |
| Diary Data | | more than 2 days per week in more than 1 week out of the |
| 1 | | first 8 weeks (Day 1 – Day 57) |
| | | Missing rescue medication (paracetamol) diary data for more |
| | | than 2 days per week in more than 1 week out of the first 8 |
| | | weeks (Day 1 – Day 57) |

<sup>\*</sup>Where medications listed above need to be identified programmatically, a list of dictionary codes from the GSK Drug dictionary will be defined with input from the study physician and coding dictionary analyst. The list will be created prior to unblinding and stored in a spreadsheet in refdata.

# 14.2. Appendix 2: Schedule of Activities

# 14.2.1. Screening

| | SCREENING PERIOD | - |
|---|---|---|
| | Screening may be performed | |
| | l | |
| PROCEDURE | across one or more visits. | NOTES |
| | Part A: up to 28 days before Day | |
| | 1. Part B: from Day -42 to Day -5 | |
| | (up to 42 days before Day 1) | |
| Informed consent | X | , |
| Inclusion and exclusion criteria | Х | |
| Demography | Х | |
| Full physical examination | X | |
| Medical/medication/drug/alcoho l history | х | |
| Alcohol and tobacco screens | х | As per standard local practice. Smoking permitted only in Part B. |
| Urine drug screen | х | |
| HIV, Hepatitis B (HBsAg and | | |
| HBcAb) and Hepatitis C (HepC | X | |
| antibody) screening | | |
| Holter monitoring | Х | 24 hour for Part B only |
| 12-lead ECG | Triplicate | , |
| Vital signs | · x | See SRM for details |
| Echocardiogram | Х | |
| Haematology, clinical chemistry, | | |
| urinalysis | X | Refer to Appendix 2. C3, C4 and BNP are included. |
| | | Documented negative COVID test within two days of |
| COVID-19 (SARS-CoV-2) | X | initial screening <u>OR</u> test performed at the time of |
| 25 (27 11.0 20 1 2) | , | initial screening |
| TB Screening (QuantiFERON) | х | militar servering |
| FSH and estradiol (in WNCBP) | X | |
| Height and weight | X | |
| Treight and weight | ^ | Inclusion Criterium. X ray performed only if ALL |
| | | · · ——— |
| V vov (KO) of index knoon init | Dowt D | other inclusion and exclusion criteria were already |
| X-ray (K&L of index knee joint) | Part B | met at initial screening (except NRS). Allow at least |
| | | 7 calendar days for the X-ray result to be returned |
| | | from central reading. |
| | | Scores will be recorded over the 7 consecutive |
| Daily pain scores (Digital Tool) | Part B (Day -7 to Day -1) | evenings preceding dosing. Average result (Baseline |
| | | value) will be evaluated for inclusion. |
| SAE assessment | Х | From signing consent |

# 14.2.2. Part A Cohorts Without Blister: 0.1 and 0.3 mg/kg IV

| | <u> </u> | | | Day | _ | _ | _ | _ | | | | Early | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | -1 | 1 | 2 | 3 | _ | 15 | 22 | 29 | 43 5 | 57 8 | 5 11 | | Allowed visit windows are detailed in the SRM |
| Out-patient visit | | | | | | | | | | | | | <sup>1</sup> Final follow-up visit for 0.1 mg/kg cohort |
| | | | | | X | Х | Х | Х | X | x x | , X | Х | <sup>2</sup> Final follow-up visit for 0.3 mg/kg cohort |
| Admission in clinical unit | Х | | | | | | | | | | t | | |
| Discharge from dinical unit | | | | X | | | | | | | т | | |
| Inclusion and exclusion criteria | X | | | | | | | | | | $\top$ | | |
| Brief physical examination | Х | Х | х | X | Х | х | х | Х | Х | x x | X | X | |
| Alcohol and tobacco screens | Х | | | | | | | | | | | | As per standard local practice |
| Urine drug screen | X | | | | | | | | | | Т | | |
| | | | | | | | | | | Т | Т | | Telemetry from at least 12 hrs before dosing until 12hrs post |
| | X | | | | | | | | | | 1 | | dose. Output to be reviewed for abnormalities prior to dosing on |
| Cardiac telemetry | | | | | | | | | | | | | Day 1. |
| | | | | | | | | | | Т | Т | | On day -1 and day 1 ECGs may be generated from telemetry |
| | Triplicate | x <sup>1</sup> | х | x | x | x | х | x | x I | x x | l <sub>x</sub> | x | On Day 1, pre dose then every 30 mins during infusion (i.e. 30 |
| | Implicate | X | ^ | ^ | l^ | ^ | ^ | ^ | ^ ' | ^ ^ | T^ | _ ^ | mins and 60mins after start of infusion) and then 1 hr post end of |
| 12-lead ECG | | | | | | | | | | | ┸ | | infusion. |
| | | | | | | | | | | | П | | On Day 1, pre dose then every 15 mins during infusion (i.e. 15, |
| | X | X1 | Х | X | Х | Х | х | х | X : | x x | X | X | 30, 45 and 60mins post the start of infusion) and then 30 mins, 1, |
| Vital signs | | | | | | | | | | | | | 2 and 4 hr post end of infusion. |
| | | | 24hr | 48hr | | П | | | $\neg$ | $\top$ | Т | | |
| | X | | post | post | Х | Х | х | х | X | Χ | X | × | |
| Haematology, clinical chemistry, urinalysis | | | dose | dose | | | | | | | ┖ | | |
| Weight | X | | | | | | | | | $\perp$ | $\perp$ | | Weight to be used to calculate the study treatment dose. |
| | | Pre- | | | | | | | | | 1 | | |
| Randomization | | dose | | | | | | | | _ | ┸ | | |
| CCI | | | | | | | | | | | | | |
| Study treatment dosing | | Х | | | | | | | | | | | |
| AE assessment | | ζ | | | | | | | | | .> | X | |
| SAE assessment | < | | | | | | | | | | > | X | |
| Concomitant medication review | < | | | | | | | | | | > | X | |

# 14.2.3. Part A Cohorts With Blister: 1 mg/kg IV

| | | | | | Day | | | | | | | | | | Early | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Proce dure | -1 | 1 | 2 | 3 | 7 | 8 | 15 | 22 | 29 | 42 | 43 | 57 | 85 | 113 | withdrawal | Allowed visit windows are detailed in the SRM |
| Out-patient visit | | | | | | | Х | х | х | | | х | х | х | × | |
| Admission in clinical unit | × | | | | Х | | | | Г | Х | | | | | | |
| Discharge from clinical unit | | | | X | | Х | | | П | | Х | | | | | |
| Inclusion and exclusion criteria | × | | | | | | | | | | | | | | | |
| Brief physical examination | × | X | × | X | х | | Х | х | × | х | | х | х | х | × | |
| Alcohol and tobacco screens | X | | | | | | | | | | | | | | | As per standard local practice |
| Urine drug screen | х | | | | | | | Г | П | | | | | | | |
| Cardiac telemetry | × | | | | | | | | | | | | | | | Telemetry from at least 12 hrs before dosing until 12hrs post dose. Review for abnormalities prior to dosing on Day 1. |
| 12-lead ECG | Triplicate | X <sup>2</sup> | х | × | x | | x | x | x | × | | x | × | x | × | On Day -1 and Day 1 ECGs may be generated from telemetry On Day 1, pre dose then every 30 mins during infusion (i.e. 30 mins and 60 mins after start of infusion) and then 1 hr post end o infusion. |
| Vital signs | × | X1 | × | × | × | | х | x | × | x | | x | × | x | × | On Day 1, pre dose then every 15 mins during infusion (i.e. 15, 30, 45 and 60mins post the start of infusion) and then 30 mins, 1, 2 and 4 hr post end of infusion. |
| Haematology, dinical chemistry, urinalysis | X | | 24hr | 48hr | Х | | Х | х | х | Х | | Х | Х | Х | X | |
| Weight | X | | | | | | | | | | | | | | | Weight to be used to calculate the study treatment dose. |
| Randomization | | Pre-<br>dose | | | | | | | | | | | | | | |
| Induction of blister | X | | | | Х | | | ᆫ | ┺ | Х | | | | _ | | |
| Aspiration of blister fluid | | X | | | | Х | | L | L | | Х | | | | | Aspiration 21 hours (+/- 3 hours) after induction of blister. |
| Blood sample for circulating immune cells | | X | | | | Х | | L | ┖ | | х | | | | | Cohort 3 only (not needed for Cohorts 1 and 2) |
| | | | 24hr | 48hr | | | | ı | ı | | Ш | Ш | | l | l | D1 Samples to be taken at |
| PK blood sample | | X | post | post | | Х | Х | Х | Х | | х | Х | Х | Х | X | IV cohorts - pre-dose, 2 hr, 4 hr, 8 hr, and 12 hr post dose |
| CCI | | | dose | dose | | | | | | | | | | | | SC cobort - pre-dose and 8 hr post dose |
| Study treatment dosing | | X | | | | | | | | | | | | | | |
| AE assessment | | | ζ | | | | | | | | | > | | | X | |
| SAE as sessment | < | | | | | | | | | | | | > | | Х | |
| Concomitant medication review | × | | | | | | | | | | | | -34 | | X | |

# 14.2.4. Part A Cohorts With Blister: 3 and 10 mg/kg IV and SC

| | | | | | | Day | | | | | | | | | Early | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | -1 | 1 | 2 | 3 | 7 | 8 | 15 | 22 | 28 2 | 29 4 | 13 5 | 7 8 | 5 11 | 3 1 | 11 withdrawa | Allowed visit windows are detailed in the SRM |
| Out-patient visit | | | | | | | x | x | | x I | П, | x x | ( x | ۱ ) | 2 X | <sup>1</sup> Final follow-up visit for 3 mg/kg IV cohort |
| Out-patient visit | | | | | | | ^ | ^ | 1 | ^ | | ^ I ^ | ` × | , | ^ | <sup>2</sup> Final follow-up visit for 10 mg/kg IV and SC cohorts |
| Admission in clinical unit | x | | | | X | | | | X | Т | Т | Т | Т | | | |
| Discharge from clinical unit | | | | Х | | Х | | | , | X | | | | | | |
| Inclusion and exclusion criteria | X | | | | | | | | | | | | | | | |
| Brief physical examination | X | X | × | X | X | | X | X | X I | X > | X ) | X X | C X | : 3 | X | |
| Alcohol and to bac co screens | X | | | | | | | $\perp$ | $\perp$ | $\perp$ | $\perp$ | $\perp$ | $\perp$ | | | As per standard local practice |
| Urine drug screen | X | | | | | | | _ | | _ | | $\perp$ | _ | | | |
| Cardiac telemetry | × | | | | | | | | | | | | Т | | | Telemetry from at least 12 hrs before dosing until 12hrs post dose. |
| Cardiac telefficity | | | | | | | $\sqcup$ | _ | _ | 4 | _ | _ | ┸ | ㅗ | | Review for abnormalities prior to dosing on Day 1. |
| | 1 | l | l . | | | | | | | | | | 1 | | | On Day -1 and Day 1 ECGs may be generated from telemetry |
| 13 land 555 | Triplicate | X <sup>1, 2</sup> | × | × | x | | x | x | x l | x l> | x , | x x | , x | ٠, | × | On Day 1, pre dose then every 30 mins during infusion (i.e. 30 mins and |
| 12-lead ECG | Triplicate | Х. | ^ | | ^ | | ^ | ^ I | ^ l' | ^ [ ' | ^ ' | ^ ^ | ` | , , | | 60mins after start of infusion) and then 1 hr post end of infusion. 2 On |
| | 1 | l | ı | l | | | | - 1 | - 1 | - | | | 1 | | 1 | Day 1, pre dose then 1 hr post injection. |
| | | | | | | | $\Box$ | $\neg$ | $\neg$ | $\top$ | o | $\top$ | ┰ | $\neg$ | _ | On Day 1, pre dose then every 15 mins during infusion (i.e. 15, 30, 45 |
| Vital signs | × | X1.2 | × | × | x | | x | x I | x ls | x l> | x ls | x I x | c x | ٠, | × | and 60mins post the start of infusion) and then 30 mins, 1, 2 and 4 hr po |
| ortal signs | 1 ^ | ^ | ^ | ^ | ^ | | ^ | ^ I | ^ ' | ^ [ ^ | ^ 1 | ^ ^ | ` ^ | . . | ` <b>.</b> ^ | end of infusion. <sup>2</sup> On Day 1, pre dose then 1 hr post injection. |
| | | | 24hr | 24hr | | - | $\vdash$ | - | - | + | + | + | + | _ | + | end of infusion. On Day 1, pre dose then 1 hr post rejection. |
| Haematology, clinical chemistry, urinalysis | X | | p.d. | p.d. | X | | X | X | x D | x > | x > | x x | C X | ( ) | X X | |
| Weight | X | | p.a. | p. a. | | Н | | - | - | + | + | + | + | | _ | Weight to be used to calculate the study treatment dose. |
| weight | _ ^ | Pre- | _ | - | | Н | $\vdash$ | - | + | + | + | + | ┰ | + | + | Weight to be used to calculate the study treatment dose. |
| Randomization | | dose | | | | | | - 1 | | - | | | | | | |
| Induction of blister | × | dose | | _ | v | Н | $\vdash$ | _ | × | + | + | + | ╈ | + | + | |
| Aspiration of blister fluid | _^ | X | _ | _ | l^ | × | $\vdash$ | _ | * | x | + | + | ╈ | + | + | Aspiration 21 hours (+/- 3 hours) after induction of blister. |
| Blood sample for circulating immune cells | | x | | | $\vdash$ | × | $\vdash$ | $\dashv$ | 1 | x I | + | + | + | - | _ | Papiration 21 riod a (4) - 3 riod a y arter induction of crister. |
| CCI | | - " | | | | - | | | | | | | | | | |
| Study treatment dosing | | X | | | | | | | т | т | Т | Т | Т | | $\overline{}$ | |
| Study treatment dosing AE assessment | | X | 6- | | | | | | | T | 1 | | Ţ | | x | |
| | | Х | | | | | | | | | | | | | × | |

#### 14.2.5. Part B

| PROCEDURE | SCREEN | | | a | TRE | ATN | ИEN | IT PE | RIO | D ( | 8 W | ks) | | | | b FC | LLOV | N-UP | (~12 | Wks) | Early | See two footnotes. NOTES a) Treatment Period = Day 1 to 57. b) Follow-Up Period = Day 57 to 141. c) Day 141 (End of Study Visit) is ~13 wks since last dose on Day 50. |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| DAY | Day -41 | 1 | 2 | 5 | 8 | 15 | 22 | 23 | 26 | 29 | 36 | 43 | 50 | 51 | 57 | 71 | 85 | 99 | 120 | c <sub>141</sub> | raw | Visit Windows: 1) Within 96 hours of Day 1 Days 15 to 71 (±1), Days 85 to 141 (±2). |
| Out-patient visit | X | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | X | X | Х | Tel. | Х | Х | Tel = telephone contact to check AEs and ConMeds (Day 120). |
| Discharge from clinical unit | | Χ¹ | | | X2 | X <sup>2</sup> | Χ² | | | Χ² | Χ² | Χ² | Χ² | | | | | | | | | <ol> <li>Day 1: Discharge <u>not</u> sooner than 4 hours post-start of SC injections.</li> <li>Remaining dosing<br/>days: discharge not sooner than 2 hours post-start SC injections.</li> </ol> |
| Inc. & Exc Criteria | Х | Х | | | | | | | | | | | | | | | | | | | | Re-check clinical status before first dose. |
| Brief Phys. Exam. | Х | (X) | Х | Χ | Χ | χ | χ | Χ | Χ | χ | Χ | Χ | Х | Χ | Х | X | Х | Х | | Х | X | |
| Alcohol and drug screen | X | Х | | | Х | Х | Х | | | Х | Х | Х | X | | Х | | | | | | | Methods as per standard local practice |
| 12-lead ECG (Triplicate) | X | (X) <sup>1</sup> | Х | | $X^1$ | $X^1$ | $X^{1}$ | | | χı | χı | Χl | Χì | | Х | X | X | | | Х | X | <ol> <li>On Dosing Days: pre-dose, and then 30 and 60 mins after post-start of dosing.</li> </ol> |
| Vital signs | Х | (X) <sup>1</sup> | х | | X <sup>2</sup> | χ² | X2 | | | χ² | χ² | χ² | X <sup>2</sup> | | Χ | х | Х | | | Х | Х | <ol> <li>Day 1: pre-dose, and then 30 mins, 1, 2, 3 and 4 hrs post-start of dosing. 2) On other dosing<br/>days: pre-dose, 1 h and 2 hrs.</li> </ol> |
| Haematology, clinical<br>chemistry, urinalysis | (X) 1,2 | | х | | Х | Х | х | | | Х | Х | Х | х | | χ² | х | х | х | | Х | х | Appendix 2. Samples taken prior to dosing, as appropriate. ADDITIONALLY: 1) Complement C & C4 (Screening only). 2) BNP (Screening & Day 57 only). |
| SARS-CoV-2 PCR<br>Mandatory | X <sup>1</sup> | | | | | | | | | | | | | | χ | | | | | Х | Х | 1) SARS-CoV-2 PCR NEGATIVE RESULT to be obtained prior to the 1st dose |
| SARS-CoV-2 PCR<br>Optional | | | | | | ←1 | | | | | ←1 | | | | | | | | | | | <ol> <li>Recommended optional SARS-CoV-2 PCR test to be obtained ideally four days before the 3<br/>and 6th dose such that a result is available prior to dosing on those days</li> </ol> |
| Daily Pain (Digital Tool) | See Screen | < | | | | | | D | aily F | Pain- | | | | | | | > | | | | | N.B. Pain recorded daily using a digital tool (Evenings of Day 1 to Day 84) |
| WOMAC | | (X) | | | Х | Х | | | | Χ | | Х | | | Х | X | X | Х | | Х | X 1 | WOMAC, PtGA (participant) & PhGA (Physician Global Assessments) completed prior to ALL |
| PtGA & PhGA | | (X) | | | Х | Х | Х | | | Х | Х | Х | Х | | Х | X | Х | Х | | Х | X 1 | other assessments and blood draws. 1) If withdrawal occurs earlier than Day 85. |
| Pain Detect (Digital Tool) | | (X) | | | | | | | | | | | | | Х | | Х | | | | Х | Perform PainDetect after completing WOMAC/Patient & Physician Global Assessment. |
| Randomization | | Х | | | | | | | $\dashv$ | | | | | | | | | $\vdash$ | - | | | |
| Dosing (SC injections) | | х | | | х | х | х | | $\neg$ | х | х | х | х | | | | | $\overline{}$ | | | | Allow at least 1 hour to thaw vials at room temp (or thaw 18 hours overnight at 2-8°C). |

All activities and blood samples are to be acquired prior to dosing (on dosing days), unless stated otherwise.

(X) denotes the Baseline Value.

Trial Questionnaire

X Optional trial-based questionnaire for participant completion.

#### 14.3. Appendix 3: Assessment Windows

Acceptable time windows around the nominal time points for specific assessments will be included in the Study Reference Manual (SRM) and assessments performed within these time windows will not constitute a protocol deviation.

The table below describes the visit days for each week (Week 1-12). All available diary data in each of the weekly intervals will be used to calculate the Average Knee Pain Intensity, Worst Knee Pain Intensity and colored for that study week.

| Study Week | Study Day | Phase |
|------------|-----------|------------|
| BL | -7 to -1 | Baseline |
| 1 | 1 to 7 | Treatment |
| 2 | 8 to 14 | Treatment |
| 3 | 15 to 21 | Treatment |
| 4 | 22 to 28 | Treatment |
| 5 | 29 to 35 | Treatment |
| 6 | 36 to 42 | Treatment |
| 7 | 43 to 49 | Treatment |
| 8 | 50 to 56 | Treatment |
| 9 | 57 to 63 | Follow-up* |
| 10 | 64 to 70 | Follow-up |
| 11 | 71 to 77 | Follow-up |
| 12 | 78 to 84 | Follow-up |

<sup>\*</sup>Follow-up here means that the participant is no longer receiving the study medication/placebo, so only for informative purposes. Participants will be considered on treatment during the whole duration of the study (20 weeks).

All other assessments will use the nominal timepoints unless otherwise specified.

# 14.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

# 14.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to the first dose.

| Study Phase | Definition |
|---------------|---------------------------------------------|
| Pre-Treatment | Date/time < Study Treatment Start Date/time |
| On-Treatment | Study Treatment Start Date ≤ Date/time |

Refer SOA in Appendix 2 for details of follow-up for each Cohort and Part.

#### 14.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is >7 days prior to first dose. |
| Concomitant | Any medication that is not a prior |

NOTE: Refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing

In addition, the following phase will also be calculated:

| Study Phase | Definition |
|---|---|
| Prohibited<br>Medication | If medication has start date on or before Day 71 and is either ongoing or has end date on or after 7 days prior to first dose (Section 6.6 of the Protocol) |
| Phase | end date on or after 7 days prior to first dose (Section 6.6 or the 1 rotocor) |

## 14.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|--------------------|------------------------------------------------|
| Treatment Emergent | If AE start date >= Study Treatment Start Date |

#### NOTES:

Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 14.5. Appendix 5: Data Display Standards & Handling Conventions

# 14.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | UK1SALX00175 |
| HARP Compound | HARP Compound \arprod\gsk3858279\mid207804 |
| Analysis Datasets | |
| Analysis datasets will be created according to Legacy GSK A&R dataset standards | |
| Generation of RTF and PDF Files | |
| RTF and PDF files will be generated. | |

#### 14.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - o 6.01 to 6.11: Principles Related to Summary Tables
  - o 7.01 to 7.13: Principles Related to Graphics
- All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology.

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DPs) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

Actual values will be used in listings. The following criteria will be used in tables and figures:

- For all Biomarkers, the following precision places will be applied:
  - Summary Statistics: 4 significant figures for Mean and Median, 5 significant figures for SD, 3 significant figures for Min and Max, in all cases but Blister Volume parameter.
  - For Blister Volume parameter: 2DP's, 3 DP's for Mean and Median, 4 DP's for SD, 3 DP's for Min and Max
- For PD endpoints, which are blinded until DBF, determination of an appropriate presentation of significant figures will be made after unblinding in line with the IDSL principles

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to the first dosing will be used in figures, summaries and planned time relative to the last dosing will be used in statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in by-visit summary tables and figures.
- All unscheduled visits will be included in listings and determination of worst-case values.

| · · | |
|---|---|
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 – do not report 95% CI unless |
| | otherwise specified. |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| D. C. L. IDOL OL C. C. L. D. C. L. Z.O.L. Z.O. | |

Refer to IDSL Statistical Principals 7.01 to 7.13.

# 14.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non- | PC WNL file (CSV format) for the non compartmental analysis by Clinical |
| Linear (WNL) File | Pharmacology Modelling and Simulation function will be created according |
| | to VQD-GUI-000722 (6.0). |
| | Note: Concentration values will be imputed as per VQD-GUI-000722 (6.0). |
| Descriptive | Refer to IDSL PK Display Standards. |
| Summary | Refer to IDSL Statistical Principle 6.06.1. |
| Statistics, | Note: Concentration values will be imputed as per VQD-GUI-000722 (6.0) |
| Graphical Displays | for descriptive summary statistics/analysis and summarized graphical |
| and Listings | displays only. |
| NONMEM/PK/TE/P | PK/TE/PD file (CSV format) for the PK/TE/PD analysis by Clinical |
| D File | Pharmacology Modelling and Simulation function will be created according |
| | to the data specification detailed in Section 11.1 Pharmacokinetic / |
| | / Pharmacodynamic Dataset Specification. |
| Pharmacokinetic Pa | rameter Derivation |
| PK Parameter to be | All PK parameters described in Section 9.1.1.2 (Part A and Part B). |
| Derived by CPMS | |
| PK Parameter to be | The following PK parameters will be derived by programmer for Part A: |
| Derived by | <ul> <li>Within subject and timepoint blister fluid: serum concentration ratio</li> </ul> |
| Programmer | for GSK3858279. |
| Pharmacokinetic Pa | rameter Data |
| Is NQ impacted PK | Yes, refer to SOP_314000. |
| Parameters Rule | |
| Being Followed | |
| Descriptive | Refer to IDSL PK Display Standards. |
| Summary | Refer to VQD-GUI-000722 (6.0). |
| Statistics, | |
| Graphical Displays | |
| and Listings | |


#### 14.6. Appendix 6: Derived and Transformed Data

#### 14.6.1. General

#### **Subject Number**

 Participants will be assigned a unique identification number: study number concatenated subject ID number. In the case of a subject being enrolled multiple times, the first subject ID number will be used. For more details, see the AR data set specifications. Listings will include both subject ID and unique subject ID.

#### Multiple measurements at one analysis time point

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Participants having both high and low values for Normal Ranges at any post-baseline visit
  for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential
  Clinical Importance summary tables.

#### Study day

- Calculated as the number of days from first dose date:
  - $\circ$  ref date = missing  $\rightarrow$  study day = missing
  - $\circ$  ref date < first dose date  $\rightarrow$  study day = ref date first dose date
  - o ref date ≥ first dose date → study day = ref date (first dose date) + 1

#### **Nominal Visit Day**

- Nominal Visit Days were updated in protocol, however some visits may be recorded under the incorrect visit number/label for Part A only:
  - Day 112 and Day 113 will be collapsed under the Nominal Visit: Day 113.
  - Day 140 and Day 141 will be collapsed under the Nominal Visit: Day 141.

#### 14.6.2. Study Population

#### Age

- Birth date will be presented in listings as 'YYYY'.
- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any participant with a missing day will have this imputed as day '15'.
  - Any participant with a missing date and month will have this imputed as '30th June'.
- Calculated based on the screening date

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

#### Race Category

- The five high level FDA race categories and designated Asian subcategories will be summarised along with all combinations of high level categories which exist in the data.
- The high level FDA race categories and designated Asian subcategories are:
  - AMERICAN INDIAN OR ALASKA NATIVE
  - ASIAN
    - CENTRAL/SOUTH ASIAN HERITAGE
    - JAPANESE HERTIAGE/EAST ASIAN HERITAGE/SOUTH EAST ASIAN HERITAGE
    - MIXED ASIAN RACE (only required if data exists)
  - BLACK OR AFRICAN AMERICAN
  - NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER
  - o WHITE
- A subject who selects a combination of races will be counted in a row within "MULTIPLE" or within the "MIXED ASIAN RACE", not in each of the constituent terms.

#### **Extent of Exposure**

- Number of days of exposure to study drug in Part B will be calculated based on the formula:
  - Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1+18\*5
  - Note: The half life of the drug is approximately 18 days. Hence 5\*18 =~ 90 days is added in the equation of duration of exposure.
- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The summary statistics based on the frequency of injections would be provided in the exposure display for Part B.

#### 14.6.3. Efficacy

#### Derivations

#### WOMAC Osteoarthritis Index

- WOMAC questionnaire covers pain, stiffness and function related to osteoarthritis in the index knee. Participants will respond to each question using an 11-point NRS (0-10), with 0=
- For each of the subscales pain, stiffness and function, the average of all the scores within
  that subscale will be calculated for each subject at each timepoint such that the average lies
  within the range of 0 to 10.
- The questions 1 to 5 constitute the subscale WOMAC pain, questions 6 and 7 constitute the subscale WOMAC stiffness, questions 8 to 24 constitute the subscale WOMAC function.
- If any of the scores within a subscale is missing for a participant, then the subscale will not be computed and will be set to missing for that participant.

# Daily Pain NRS

- Average knee pain intensity: mean over the 7 days prior to each assessment visit
- Worst knee pain intensity: mean over the 7 days prior to each assessment visit

#### 14.6.4. Safety

#### **ECG Parameters**

#### **RR Interval**

- IF RR interval (msec) is not provided directly, then RR can be derived as:
  - [1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

- if both the QTcB and QTcF values are machine read and provided, RR will not be calculated.
- If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value, THEN do not derive.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as:

$$QTcB = \frac{\dot{Q}T}{\sqrt{\frac{RR}{1000}}} \qquad \qquad QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### **Worst Case Rules**

Worst case finding based on the interpretation and the clinical significance:

- Count the subject as 'ABNORMAL' and 'CLINICALLY SIGNIFICANT', if any of the findings are 'ABNORMAL' and 'CLINICALLY SIGNIFICANT' during the time period/Post-Baseline.
- Else count the subject as 'ABNORMAL' and 'NOT CLINICALLY SIGNIFICANT', if any of the findings are 'ABNORMAL' and 'NOT CLINICALLY SIGNIFICANT' and none of the findings are 'ABNORMAL' and 'CLINICALLY SIGNIFICANT' during the time period/Post-Baseline.
- Else count the subject as 'NORMAL' if there is a finding of 'NORMAL' and none of the findings are 'ABNORMAL during the time period/Post-Baseline.
- Otherwise, do not count the subject during the time period/Post-Baseline, i.e. little n will reflect that the subject is not counted in the time period/Post-Baseline..

#### **Laboratory Parameters**

- All BLQ values will be imputed with ½ LLOQ.
- All ALQ values will be imputed with the ALQ + [smallest positive number with the same number of decimal places as the ALQ is reported with]
- Values reported as < x are assumed to have an LLOQ of x.</li>
- Values reported as > x are assumed to have an ALQ of x.

## 14.6.5. Immunogenicity

A seed (5315) will be generated using code as outlined in Section 14.9.2. This will be saved in the refdata area.

- Using the generated seed, random numbers will be generated for all subjects that exist in the imgen dataset.
- These subjects will be ordered based on the random number and letters assigned sequentially (i.e. the patient with the smallest random number was 'a', the next patient 'b' and so on).

# 14.7. Appendix 7: Reporting Standards for Missing Data

# 14.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>A participant is considered to have completed the study if he/she has completed all phases of the study including the final follow-up visit</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 14.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to |
| | blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant</li> </ul> |
| | listing displays. Unless all data for a specific visit are missing in which |
| | case the data is excluded from the table. |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not</li> </ul> |
| | considered to be missing data and should be displayed as such. |

# 14.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Partial dates will be displayed as captured in participant listing displays.</li> <li>Where necessary, display macros may impute dates as temporary variables for sorting data in listings only. In addition, partial dates may be imputed for 'slotting' data to study or for specific analysis purposes.</li> </ul> |
| Adverse<br>Events | <ul> <li>Imputations in the adverse events dataset are used for slotting events to the appropriate study time periods and for sorting in data listings.</li> <li>Partial dates for AE recorded in the CRF will be imputed using the following conventions:</li> <li>Missing start day</li> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = 1st of month.</li> <li>Else if study treatment start date is not missing: <ul> <li>If month and year of start date = month and year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = 1st of month.</li> <li>Else set start date = study treatment</li> </ul> </li> </ul> |
| | start date. o Else set start date = 1st of month. |

| | Reporting Detail | |
|---|---|---|
| | Missing start day and month | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = January 1.</li> <li>Else if study treatment start date is not missing: <ul> <li>If year of start date = year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start date = January 1.</li> <li>Else set start date = study treatment start date.</li> <li>Else set start date = January 1.</li> </ul> </li> </ul> |
| | Missing stop day | Last day of the month will be used. |
| | Missing stop day and month | No Imputation |
| | Completely missing start/end date | No imputation |
| Concomitant<br>Medications | | r any concomitant medications recorded in the CRF will be the following convention: |
| | | <ul> <li>If study treatment start date is missing (i.e. participant did not start study treatment), then set start date = 1st of month.</li> <li>Else if study treatment start date is not missing: <ul> <li>If month and year of start date = month and year of study treatment start date then</li> <li>If stop date contains a full date and stop date is earlier than study treatment start date then set start</li> </ul> </li> </ul> |
| | | not start study treatment), then set start date = 1st of month. • Else if study treatment start date is not missing: o If month and year of start date = month and year of study treatment start date then • If stop date contains a full date and stop date is earlier than study |
| | Missing start day and month | not start study treatment), then set start date = 1st of month. • Else if study treatment start date is not missing: o If month and year of start date = month and year of study treatment start date then • If stop date contains a full date and stop date is earlier than study treatment start date then set start date= 1st of month. • Else set start date = study treatment start date. |


| Element | Reporting Detail |
|---|---|
| | Missing end day and A '31' will be used for the day and 'Dec' will be used for the month. |
| | Completely missing start/end date |
| | The recorded partial date will be displayed in listings. |

# 14.8. Appendix 8: Values of Potential Clinical Importance

# 14.8.1. PCI Values for Part A

# 14.8.1.1. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | Bpm | < 40 | > 110 |

# 14.8.1.2. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | Ratio of | Male | 0.39 | 0.54 |
| Hematocrit | 1 | Female | 0.35 | 0.49 |
| | I | $\Delta$ from BL | ↓0.075 | |
| | a/I | Male | 124 | 180 |
| Hemoglobin | g/L | Female | 109 | 180 |
| | | $\Delta$ from BL | <b>↓25</b> | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.75 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x109/ L | | 100 | 550 |
| White Blood Cell Count (WBC) | x109/ L | | 2.5 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | | | 1.3 X ULN |
| Creatinine | umol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO <sub>2</sub> | mmol/L | | 18 | 32 |
| Creatinine Kinase | mg/dL | | | >1.6 X ULN |
| C-reactive Protein | mg/L | | | ≥3.0 |
| Troponin T | ng/L | | | 14.1 |

| Liver Function | | | |
|---|---|---|---|
| Test Analyte | Units Category Clinical Concern Range | | Clinical Concern Range |
| ALT/SGPT | IU/L | High | ≥2xULN |
| AST/SGOT | IU/L | High | ≥2xULN |
| AlkPhos | IU/L | High | ≥2xULN |
| T Bilirubin | µmol/L | High | ≥1.5xULN |
| T. Bilirubin + ALT | µmol/L<br>IU/L | High | ALT≥3xULN AND bilirubin≥ 1.5xULN |

# 14.8.1.3. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | >500 |
| Absolute PR Interval | msec | <110 | >220 |
| Absolute QRS Interval | msec | <75 | >120 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | >60 |

# 14.8.2. PCI Values for Part B

# 14.8.2.1. Vital Signs

| Vital Sign Parameter | Units | Clinical Concer | Clinical Concern Range |
|---|---|---|---|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

# 14.8.2.2. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | Datio of | Male | 0.39 | 0.54 |
| Hematocrit | Ratio of | Female | 0.35 | 0.49 |
| | I | $\Delta$ from BL | ↓0.075 | |
| | g/L | Male | 124 | 180 |
| Hemoglobin | | Female | 109 | 180 |
| | | $\Delta$ from BL | <b>↓25</b> | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.75 | 4.5 |
| Neutrophil Count | x109/ L | | 1.5 | 8.0 |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| White Blood Cell Count (WBC) | x109/ L | | 2.5 | 15 |

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Category Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Clinical Chemistry | | | | |
| Laboratory Parameter | Units | Category | Clinical Concerr | n Range |
| | | | Low Flag (< x) | High Flag (>x) |
| Calcium | mmol/L | | 2 | 2.60 |
| Creatinine | umol/L | Male | | 120 |
| | | Female | | 100 |
| Creatinine | umol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 8 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Troponin T | ng/L | | | 14.1 |
| NT-pro BNP | ng/L | | | 125.2 |

| Liver Function | | | |
|---|---|---|---|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | IU/L | High | ≥1.5xULN |
| AST/SGOT | IU/L | High | ≥1.5xULN |
| AlkPhos | IU/L | High | ≥1.5xULN |
| T Bilirubin | µmol/L | High | ≥1.5xULN |
| T. Bilirubin + ALT | µmol/L | Lligh | ALT≥3xULN AND bilirubin≥ 1.5xULN |
| I. BIIIIUDIII + AL I | IU/L | High | ALTEGROLIN AND DIIIIUDIIIE 1.5XULIN |

| Immunology | | | | |
|---|---|---|---|---|
| Toot Analyte | Units | Category | Clinical Concern Range | |
| Test Analyte | | | Low Flag ( <x)< th=""><th>High Flag (&gt;x)</th></x)<> | High Flag (>x) |
| Complement C3 | g/L | High | 0.85 | 1.8 |
| Complement C4 | g/L | High | 0.1 | 0.4 |

| Virology | | | |
|----------------------|-------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| Hepatitis C Antibody | N/A | High | Reactive |

# 14.8.2.3. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | <350 | >450 |
| Absolute PR Interval | msec | <110 | >220 |
| Absolute QRS Interval | msec | <75 | >120 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | >50 |

#### 14.9. Appendix 9: Statistical Algorithms and Model Checking

#### 14.9.1. Calculation of SD from Bayesian Repeated Measures model

1. Calculate the R Correlation matrix (correlation matrix for the repeated measures [in this case visit])

$$R_{corr} = \begin{bmatrix} 1 & \rho_{1,2} & \dots & \rho_{1,8} \\ & 1 & \dots & \rho_{2,8} \\ & & \dots & \dots \\ & & & 1 \end{bmatrix}$$

2. Calculate the number of subject contributing data up to each week (e.g. 32 subjects have up to week 8, a further 4 subjects contribute up to week 6 only, 3 more contribute data up to week 4 only.

$$m{n}_{cont} = egin{bmatrix} n_{1,8} \\ n_{2,8} \\ ... \\ n_{7,8} \end{bmatrix} = egin{bmatrix} n_1 \\ n_2 \\ ... \\ n_7 \end{bmatrix} - egin{bmatrix} n_8 \\ n_8 \\ ... \\ n_8 \end{bmatrix}$$

$$ESS_8 = n_8 + \sum_{i=1,...7} \rho_{i,8} n_{i,8}$$

3. Calculate the SD

$$SD_{estimate,8} = SE_8 * \sqrt{ESS_8}$$

## 14.9.2. Model Checking & Diagnostics

#### **Bayesian Repeated Measures Model**

Seeds for all planned analyses will be determined using the following SAS code

data temp;

do i=1 to #seed;

number=round(10000\*ranuni(207804),1); output;

end;

run;

The following points are for guidance and illustration and do not guarantee a successful model convergence. They cannot cover all eventualities and do not remove the requirement to do what is best for the specific set of observed data being modelled.

#### **Priors**

Unless otherwise specified the following would be the default approach to selecting prior distributions:

 Vague priors of the form Normal(0, Var=1E6) would be assigned to each fixed effect in the proposed statistical model.

- Vague Inverse-gamma priors of the form IGamma(0.001,0.001) would be assigned to standalone variance parameters that are not expected to take values near zero (e.g. for the residual variance rather than a random effect variance component)
- For stand-alone variance parameters that may take values close to zero a noninformative prior of the form Uniform(0, XXX) may be assigned for the SD
- For repeated measures models Inverse-Wishart priors will be assigned for the Variance Covariance matrix (VCV). They would use degrees of freedom equal to the dimension of the VCV matrix and an Identity matrix (of the same dimension).
  - If there are issues with those variance parameters then the Identitity matrix may be replaced with a diagonal matrix that uses best guesses for the residual variance at each repeated measure time point (or the residual estimates from fitting simple models).
  - It is good practice to ensure that each prior distribution is visualised to ensure it appears sensible and allows clinically plausible response values, whilst not allowing impossible values to be drawn with high probability and that if it is intended to be non-informative it is doing so over the region of the likelihood function.

#### Checking convergence and other diagnostics

The key model diagnostic output is the MCSE/SD ratio for each parameter:

- Adequate values for the number of MCMC samples / thinning / number of burn in samples should be chosen to ensure that the MCSE/SD for the key parameters is below 0.01 (e.g. key parameters those associated with treatment, or as pre-specified comparisons of interest) in each final model.
- For other model parameters, try to get the MCSE/SD values as close to 0.01 as possible, but if there is significant autocorrelation then values below 0.05 would be considered acceptable.
- In addition, the number of tuning units and maximum number of tuning iterations may be increased to find a better multivariate normal approximation to the parameters, which in turn may reduce the MCSE/SD values
- Where possible the code should be written to allow the SAS compiler to identify and use conjugate sampling, since this can greatly reduce the corresponding MCSE/SD values
- Models selected with MCSE/SD values above 0.01 (for key parameters) or 0.05(for other parameters) would need a brief remark/justification added to the CSR to clarify why it was not possible to reach the targets and why it is believed the subsequent model still has utility.

Use of the default SAS PROC MCMC diagnostic plots should be made and where possible:

- Autocorrelation should decline rapidly and show no oscillation patterns
- Worm plots should show the chain appears to be stationary and mixing, i.e.
  - o Constant mean, constant variance
  - Moving around the parameter space freely (not getting "stuck" at similar values for a large number of iterations before moving on again)
  - Moving rapidly between extremes
  - The posterior density should look reasonable for each parameter (e.g. for posterior parameters expected to follow a normal distribution the density plot should not
- appear bi-modal, but for parameters acting as binary flags then bi-modal is acceptable)
- Correlation structures between relevant posterior parameters (and/or parameters in each PARMS block) should be explored using graphical methods. This can provide information about what potential issues may be and also what corrective action(s) may be worthwhile attempting.

# 14.10. Appendix 10: Abbreviations & Trade Marks

## 14.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| AUC | Area Under the Concentration-Time Curve |
| A&R | Analysis and Reporting |
| BNP | N-terminal pro B-type natriuretic peptide |
| BUN | Blood urea nitrogen |
| CI | Confidence Interval |
| Cmax | Maximum observed concentration |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> /CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DEC | Dose Escalation Committee |
| DEP | Dose Escalation Plan |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure |
| | Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| MCH | Mean Corpuscular Hemoglobin |
| MCV | Mean Corpuscular Volume |
| OA | Osteoarthritis |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PhGA | Physician Global Assessment |
| PK | Pharmacokinetics |
| PP | Per Protocol |
| CCI | |

| Abbreviation | Description |
|--------------|--------------------------------------------------------|
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| RBC | Red Blood Cell Count |
| SAC | Statistical Analysis Complete |
| SOA | Schedule of Activities |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TLF | Tables, Listings and Figures |
| WBC | Whole Blood Count |
| WOMAC | Western Ontario & McMaster Universities Osteoarthritis |
| | Index |

### 14.10.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| None |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| WinNonlin |
| SAS |
| NONMEM |

## 14.11. Appendix 11: List of Data Displays

## 14.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | | Figures | |
|---|---|---|---|---|
| | Part A | Part B | Part A | Part B |
| Safety Review | N/A | 1 | N/A | N/A |
| Sample Size Re-estimation | N/A | 2 | N/A | N/A |
| Study Population | 1.01 to 1.09 | 1.10 to 1.28 | N/A | N/A |
| Safety | 2.01 to 2.16 | 2.17 to 2.39 | N/A | N/A |
| Pharmacokinetic | 3.01 to 3.06 | 3.07 to 3.08 | 3.01 to 3.06 | 3.07 to 3.09 |
| Pharmacodynamic | 4.01 to 4.05 | 4.06 to 4.08 | 4.01 to 4.03 | 4.04 to 4.06 |
| CCI | | | | |
| Efficacy | N/A | 6.01 to 6.21 | N/A | 6.01 to 6.15 |

| Section | Listings | |
|----------------|-------------------|--------------|
| | Part A | Part B |
| ICH Listings | 1 to 31, 64 to 65 | 32 to 63, 66 |
| Other Listings | 67 to 76 | 77 to 87 |

### 14.11.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated in a separate TFL Shells document.

| Section | Figure | Table | Listing |
|---------------------------|--------|---------|---------|
| Safety Review | | SR_Tn | |
| Sample Size Re-estimation | | SSR_Tn | |
| Study Population | | | |
| Safety | | SAFE_Tn | |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamic | | PD_Tn | |
| CCI | | | |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |

#### 14.11.3. Deliverables

| Delivery | Description |
|------------|--------------------------------------------|
| Part A SAC | Part A Final Statistical Analysis Complete |
| Part B SR1 | Safety Review 1 |
| Part B SR2 | Safety Review 2 |
| Part B IA1 | Interim Analysis 1 |
| Part B IA2 | Interim Analysis 2 |
| Part B IA3 | Interim Analysis 3 |
| Part B IA4 | Interim Analysis 4 |
| Part B SAC | Part B Final Statistical Analysis Complete |

# 14.11.4. Safety Review Table

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Immun | Immunogenicity – Part B | | | | |
| 1. | Safety | SR1 | Part B: Summary of Immunogenicity | | SR1, SR2 |

# 14.11.5. Sample Size Re-estimation table

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Sample | Sample Size Re-estimation – Part B | | | | |
| 2. | Safety | SSR_1 | Part B: Summary of Sample Size Re-estimation | | IA2 |

# 14.11.6. Study Population Tables

## 14.11.6.1. Part A

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Subje | Subject Disposition | | | | |
| 1.01. | Randomized | ES1 | Part A: Summary of Subject Disposition for the Subject Conclusion Record | ICH E3, FDAAA, EudraCT | Part A SAC |
| 1.02. | Screened | ES6 | Part A: Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | Part A SAC |
| Protoc | col Deviation | 1 | | | |
| 1.03. | Randomized | DV1 | Part A: Summary of Important Protocol Deviations | ICH E3 | Part A SAC |
| Popul | ation Analysed | | | | |
| 1.04. | Screened | SP1 | Part A: Summary of Study Populations | IDSL. Include footnote with population definitions. | Part A SAC |
| Demo | graphic and Bas | eline Characte | eristics | | |
| 1.05. | Randomized | DM1 | Part A: Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | Part A SAC |
| 1.06. | Enrolled | DM11 | Part A: Summary of Age Ranges | EudraCT | Part A SAC |
| 1.07. | Randomized | DM5 | Part A: Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | Part A SAC |
| Prior a | and Concomitant | t Medications | | | |
| 1.08. | Safety | CM1 | Part A: Summary of Prior Medications | ICH E3 | Part A SAC |
| 1.09. | Safety | CM1 | Part A: Summary of Concomitant Medications | ICH E3 | Part A SAC |

#### 14.11.6.2. Part B

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Subjec | t Disposition | • | | | • |
| 1.10. | Randomized | ES1 | Part B: Summary of Subject Disposition for the Subject Conclusion Record | | IA1, IA2, IA3,<br>IA4, Part B<br>SAC |
| 1.11. | Randomized | SD1 | Part B: Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | | IA1, IA2, IA3,<br>IA4,<br>Part B SAC |
| 1.12. | Screened | ES6 | Part B: Summary of Screening Status and Reasons for<br>Screen Failure | | Part B SAC |
| 1.13. | Enrolled | NS1 | Part B: Summary of Number of Subjects by Country and Site ID | | Part B SAC |
| COVID | -19 | • | | | |
| 1.14. | Randomized | PAN1A | Part B: COVID-19 Case Diagnosis Events | | Part B SAC |
| Protoc | ol Deviation | | | | |
| 1.15. | Randomized | DV1 | Part B: Summary of Important Protocol Deviations | | Part B SAC |
| Popula | tion Analysed | | | | |
| 1.16. | Screened | SP1 | Part B: Summary of Study Populations | Include footnote with population definitions. | Part B SAC |
| Demog | graphic and Base | eline Characte | eristics | | |
| 1.17. | Randomized | DM1 | Part B: Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT<br>Include KL scores | IA1, IA2, IA3,<br>IA4, Part B<br>SAC |
| 1.18. | Randomized | POP_T1 | Part B: Summary of Baseline Efficacy Parameters | Include Average & Worst Knee Pain Intensity, WOMAC, and Pain Detect | IA1, IA2, IA3,<br>IA4, Part B<br>SAC |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| 1.19. | Enrolled | DM11 | Part B: Summary of Age Ranges | EudraCT | Part B SAC |
| 1.20. | Randomized | DM5 | Part B: Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | Part B SAC |
| Medic | al Conditions | • | • | • | |
| 1.21. | Randomized | MH4 | Part B: Summary of Past Medical Conditions | ICH E3 | Part B SAC |
| 1.22. | Randomized | MH4 | Part B: Summary of Current Medical Conditions | ICH E3 | Part B SAC |
| Prior a | and Concomitan | t Medications | | • | |
| 1.23. | Safety | CM1 | Part B: Summary of Prior Medications | ICH E3 | Part B SAC |
| 1.24. | Safety | CM1 | Part B: Summary of Concomitant Medications | ICH E3 | Part B SAC |
| 1.25. | Safety | CM1 | Part B: Summary of Prior Osteoarthritis Medications | OA meds are captured on a specific CRF page | Part B SAC |
| 1.26. | Safety | CM1 | Part B: Summary of Osteoarthritis Concomitant Medications during Prohibited Medication Phase | | Part B SAC |
| 1.27. | Safety | CM1 | Part B: Summary of Osteoarthritis Concomitant Medications | | Part B SAC |
| Expos | ure | | | • | |
| 1.28. | Safety | EX1 | Part B: Summary of Exposure to Study Treatment | Provide statistics for the categories by number of injections received (4 injections, ≤ 3 injections) | Part B SAC |

# 14.11.7. Safety Tables

### 14.11.7.1. Part A

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Adver | dverse Events (AEs) | | | | |
| 2.01. | Safety | AE1CP | Part A: Summary of All Adverse Events by System Organ Class and Preferred Term | | Part A SAC |
| 2.02. | Safety | AE5A | Part A: Summary of All Adverse Events by System Organ Class and Preferred Term and Maximum Intensity | | Part A SAC |
| 2.03. | Safety | AE5A | Part A: Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity | | Part A SAC |
| 2.04. | Safety | AE15 | Part A: Summary of All Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | Part A SAC |
| Vital S | igns | | | | |
| 2.05. | Safety | VS1 | Part A: Summary of Change from Baseline in Vital Signs | Includes Baseline values. | Part A SAC |
| 2.06. | Safety | VS7 | Part A: Summary of Worst Case Vital Signs Results by PCI Criteria Post-Baseline Relative to Baseline | Include all assessments post-<br>baseline | Part A SAC |
| Labora | atory: Hematol | ogy | | | |
| 2.07. | Safety | LB1 | Part A: Summary of Hematology Changes from Baseline | Includes baseline values. | Part A SAC |
| 2.08. | Safety | LB17 | Part A: Summary of Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline | Include all assessments post-<br>baseline | Part A SAC |
| Labora | atory: Chemist | ry | | | |
| 2.09. | Safety | LB1 | Part A: Summary of Chemistry Changes from Baseline | ICH E3 | Part A SAC |
| 2.10. | Safety | LB17 | Part A: Summary of Worst Case Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline | ICH E3<br>Include all assessments post-<br>baseline | Part A SAC |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Labor | atory: Urinalys | is | | | |
| 2.11. | Safety | UR1 | Part A: Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline | | Part A SAC |
| ECG | | | | | |
| 2.12. | Safety | EG1 | Part A: Summary of ECG Findings | | Part A SAC |
| 2.13. | Safety | EG10 | Part A: Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | Use QTcB and QTcF intervals | Part A SAC |
| 2.14. | Safety | EG2 | Part A: Summary of Change from Baseline in ECG Values by Visit | Use QTcB and QTcF intervals | Part A SAC |
| 2.15. | Safety | EG11 | Part A: Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category | Use QTcB and QTcF intervals | Part A SAC |
| Telem | etry – Part A | | | | |
| 2.16. | Safety | EG1 | Part A: Summary of Telemetry Findings | | Part A SAC |

#### 14.11.7.2. Part B

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Adver | se Events (AEs | s) – Part B | | | |
| 2.17. | Safety | CP_AE1p | Part B: Summary of All Adverse Events by System Organ Class and Preferred Term | | IA3, Part B<br>SAC |
| 2.18. | Safety | AE5A | Part B: Summary of All Adverse Events by System Organ Class and Preferred Term and Maximum Intensity | | IA3, Part B<br>SAC |
| 2.19. | Safety | AE3 | Part B: Summary of Common (≥5%) Adverse Events by<br>Overall Frequency | | Part B SAC |
| 2.20. | Safety | AE5A | Part B: Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity | Include Total column. | IA3, Part B<br>SAC |
| 2.21. | Safety | AE15 | Part B: Summary of All Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | IA3, Part B<br>SAC |
| 2.22. | Safety | AE15 | Part B: Summary of Common (≥5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | Part B SAC |
| Seriou | is and Other Si | gnificant Adv | rerse Events | | |
| 2.23. | Safety | AE16 | Part B: Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | IA3, Part B<br>SAC |
| 2.24. | Safety | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | | IA3, Part B<br>SAC |
| 2.25. | Safety | AE3 | Summary of Serious Drug-Related Adverse Events by Overall Frequency | | IA3, Part B<br>SAC |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Vital S | Signs | | | | • |
| 2.26. | Safety | VS1 | Part B: Summary of Change from Baseline in Vital Signs | Include Baseline | IA3, Part B<br>SAC |
| 2.27. | Safety | VS7 | Part B: Summary of Worst Case Vital Signs Results by PCI Criteria Post-Baseline Relative to Baseline | | IA3, Part B<br>SAC |
| Labor | atory: Hematol | ogy | | | 1 |
| 2.28. | Safety | LB1 | Part B: Summary of Hematology Changes from Baseline | Include Baseline | IA3, Part B<br>SAC |
| 2.29. | Safety | LB17 | Part B: Summary of Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline | | IA3, Part B<br>SAC |
| Labor | atory: Chemist | ry | | | • |
| 2.30. | Safety | LB1 | Part B: Summary of Chemistry Changes from Baseline | | IA3, Part B<br>SAC |
| 2.31. | Safety | LB17 | Part B: Summary of Worst Case Chemistry Results by PCI Criteria Post-Baseline Relative to Baseline | | IA3, Part B<br>SAC |
| Labor | atory: Urinalys | is | | | 1 |
| 2.32. | Safety | UR1 | Part B: Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline | | IA3, Part B<br>SAC |
| ECG | | | | | _ |
| 2.33. | Safety | EG1 | Part B: Summary of ECG Findings | | IA3, Part B<br>SAC |
| 2.34. | Safety | EG10 | Part B: Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | Use QTcB and QTcF intervals | IA3, Part B<br>SAC |
| 2.35. | Safety | EG2 | Part B: Summary of Change from Baseline in ECG Values by Visit | Use QTcB and QTcF intervals | IA3, Part B<br>SAC |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| 2.36. | Safety | EG11 | Part B: Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category | Use QTcB and QTcF intervals | IA3, Part B<br>SAC |
| Immu | nogenicity | | | | |
| 2.37. | Safety | AE1CP | Part B: Summary of Treatment-Emergent Adverse Events by Highest Post-Baseline ADA Result | Split table by Positive/ Negative ADA status | Part B SAC |
| Injecti | on Site Reaction | ons | | | |
| 2.38. | Safety | SAFE_T1 | Part B: Summary of Injection Site Reactions as per specified AE Term list | Safety to provide list of HLT / Preferred Terms. Add a footnote explaining that this table was created using a pre-specified subset of MedDra AE Terms | Part B SAC |
| 2.39. | Safety | ESI1 | Part B: Summary of Characteristics of Injection Site Reactions as per specified AE Term list | Safety to provide list of HLT / Preferred Terms. Add a footnote explaining that this table was created using a pre-specified subset of MedDra AETerms | Part B SAC |

### 14.11.8. Pharmacokinetic Tables

### 14.11.8.1. Part A

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Serum | GSK3858279 | | | | |
| 3.01. | PK | PK01 | Part A: Summary of Serum GSK3858279 Concentration-<br>Time Data (ng/mL) | Please only present the median, min, max, sd (log), geometric mean and 95% CI, back-transformed from the loge scale. | Part A SAC |
| 3.02. | PK | PK06 | Part A: Summary of Derived Serum GSK3858279 Pharmacokinetic Parameters (non-transformed and log-transformed) | Include Cmax, tmax, AUC(0-t), AUC(0-∞), t½, CL, Vss. Please note that tmax should not be loge-transformed and 95% CI should not be presented. Please add the following footnote: CL= systemic clearance for IV, apparent systemic clearance for SC. | Part A SAC |
| 3.03. | PK | PK_T1 | Part A: Summary of Serum GSK3858279 Pharmacokinetic Dose Proportionality | | Part A SAC |
| 3.04. | PK | PK_T2 | Part A: Summary of SC:IV GSK3858279 Pharmacokinetic Comparison | | Part A SAC |
| Bliste | GSK3858279 | | | | |




#### 14.11.8.2. Part B



# 14.11.9. Pharmacokinetic Figures

### 14.11.9.1. Part A

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Serui | m GSK3858279 | | | | |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| 3.02. | PK | PK17 | Part A: Mean Serum GSK3858279 Concentration-Time Plots (Linear and Semi-log) | Add the following footnotes: Note: LLOQ=100 ng/mL. Note: Concentrations below LLOQ have been set to zero and included in the summary statistic calculations. Note: Any single mid-profile non-quantifiable (NQ) concentrations have been omitted. Note: Zero concentration values have been set to missing in the log-linear plot. Note: Samples have been excluded where results were missing or quantifiable pre- dose concentrations. | Part A SAC |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| 3.03. | PK | PK18 | Part A: Median Serum GSK3858279 Concentration-Time Plots (Linear and Semi-log) | Add the following footnotes: Note: LLOQ=100 ng/mL. Note: Concentrations below LLOQ have been set to zero and included in the summary statistic calculations. Note: Any single mid-profile non-quantifiable (NQ) concentrations have been omitted. Note: Zero concentration values have been set to missing in the log-linear plot. Note: Samples have been excluded where results were missing or quantifiable pre- dose concentrations. | Part A SAC |



| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| CCI | | | | | |


| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| CCI | | | | | |

#### 14.11.9.2. Part B





| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| CCI | | | | | |

# 14.11.10. Pharmacodynamic Tables

### 14.11.10.1. Part A

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Seru | erum Target Engagement | | | | |
| 4.01. | Safety | PD_T1 | Part A:<br>Summary of<br>Free & Total<br>CCL17 in<br>Serum<br>Concentration-<br>Time Data<br>(pg/mL) | Please only present the median, min, max, sd (log), geometric mean and 95% CI back-transformed from the loge scale. Apply logit transformation for % reduction parameter and present median, min, max, sd (logit), geometric mean and 95% CI, back-transformed from the logit scale. If % reduction ≤0, set to 0.1. If % reduction ≥100, set to 99.9. These imputations are needed for logit transformation. Use Student's t-distribution for CI. Add the following footnotes: Note: Free CCL17 values below the LLOQ have been imputed to ½* LLOQ. Total CCL17 values below the LLOQ whilst missing baseline values have been imputed to the median of the non-missing baseline values. Note: Free CCL17 and Total CCL17 exceeding the upper limit of quantification (ULOQ) have been excluded from the summary statistics (ULOQ Free CCL17: 3600 pg/mL, ULOQ Total CCL17: 50000 pg/mL). Note: If more than 30% of values have been imputed at any timepoint for a treatment group, then the standard deviation is not displayed. Note: Percentage reduction values <= 0 are imputed to be 0.1 and values >= 100 are imputed to be 99.9. Note: The percentage reduction parameter was logit transformed, summarised, and back-transformed using the logistic function to obtain the geometric summary statistics. The 95% CI of the geometric mean was calculated using Student's t distribution. | Part A SAC |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| 4.02. | Safety | PD_T2 | Part A: Summary of Derived Free and Total CCL17 in Serum Target Engagement Parameters (non- transformed and log- transformed) | Please only present the median, min, max, sd (log), geometric mean and 95% CI back-transformed from the loge scale. Please note that tmax and tmin should not be loge-transformed and 95% CI should not be presented. Apply logit transformation for maximum % reduction parameter and present median, min, max, sd (logit), geometric mean and 95% CI back-transformed from the logit scale. If maximum % reduction ≤0, set to 0.1. If maximum % reduction ≥100, set to 99.9. These imputations are needed for logit transformation. Use Student's t-distribution for CI. Add the following footnote: Note: Percentage reduction values <= 0 are imputed to be 0.1 and values >= 100 are imputed to be 99.9. Note: The maximum percentage reduction parameter was logit transformed, summarised, and back-transformed using the logistic function to obtain the geometric summary statistics. The 95% CI of the geometric mean was calculated using Student's t distribution. | Part A SAC |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Blist | er Target Eng | agement | | | |
| | Blister | PD_T1 | Part A:<br>Summary of<br>Free & Total<br>CCL17 in<br>Blister Fluid<br>Concentration-<br>Time Data<br>(pg/mL) | Please only present the median, min, max, sd (log), geometric mean and 95% CI back-transformed from the loge scale. Apply logit transformation for % reduction parameter and present median, min, max, sd (logit), geometric mean and 95% CI back-transformed from the logit scale. If % reduction ≤0, set to 0.1. If % reduction ≥100, set to 99.9. These imputations are needed for logit transformation. Use Student's t-distribution for CI. Add the following footnotes: Note: Free CCL17 values below the LLOQ have been imputed to ½*LLOQ. Total CCL17 values below the LLOQ have been imputed to 0. Values equal to zero at baseline have been imputed to LLOQ whilst missing baseline values have been imputed to the median of the non-missing baseline values. Note: Free CCL17 and Total CCL17 exceeding the upper limit of quantification (ULOQ) have been excluded from the summary statistics (ULOQ Free CCL17: 3600 pg/mL, ULOQ Total CCL17: 50000 pg/mL). Note: If more than 30% of values have been imputed at any timepoint for a treatment group, then the standard deviation is not displayed. Note: Percentage reduction values <= 0 are imputed to be 0.1 and values >= 100 are imputed to be 99.9. Note: The percentage reduction parameter was logit transformed, summarised, and back-transformed using the logistic function to obtain the geometric summary statistics. The 95% CI of the geometric mean was calculated using Student's t distribution. | Part A SAC |
| 4.04. | Blister | PD_T1 | Part A:<br>Summary of<br>Derived Blister | Please only present the median, min, max, sd (log), geometric mean and 95% CI back-transformed from the loge scale. Apply logit transformation for % reduction parameter and present median, min, max, | Part A SAC |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| | | | Fluid:Serum Free & Total CCL17 concentration ratio | sd (logit), geometric mean and 95% CI back-transformed from the logit scale. If % reduction ≤0, set to 0.1. If % reduction ≥100, set to 99.9. These imputations are needed for logit transformation. Use Student's t-distribution for CI. Please only present the median, min, max, sd (log), geometric mean and 95% CI back-transformed from the loge scale. Apply logit transformation for % reduction parameter and present median, min, max, sd (logit), geometric mean and 95% CI back-transformed from the logit scale. If % reduction ≤0, set to 0.1. If % reduction ≥100, set to 99.9. These imputations are needed for logit transformation. Use Student's t-distribution for CI. Add the following footnotes: Note: Free CCL17 values below the LLOQ have been imputed to ½*LLOQ. Total CCL17 values below the LLOQ have been imputed to 0. Values equal to zero at baseline have been imputed to LLOQ whilst missing baseline values have been imputed to the median of the non-missing baseline values. Note: Free CCL17 and Total CCL17 exceeding the upper limit of quantification (ULOQ) have been excluded from the summary statistics (ULOQ Free CCL17: 3600 pg/mL, ULOQ Total CCL17: 50000 pg/mL). Note: If more than 30% of values have been imputed at any timepoint for a treatment group, then the standard deviation is not displayed. Note: Percentage reduction values <= 0 are imputed to be 0.1 and values >= 100 are imputed to be 99.9. Note: The percentage reduction parameter was logit transformed, summarised, and back-transformed using the logistic function to obtain the geometric summary statistics. The 95% CI of the geometric mean was calculated using Student's t | |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| | | | | distribution. | |
| lmm | unogenicity | | | | |
| 4.05. | Safety | IMM1 | Part A:<br>Summary of<br>Immunogenicity | | Part A SAC |

### 14.11.10.2. Part B

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Seru | Serum Target Engagement | | | | |

| 4.06 | . Safety | PD_T1 | Part B:<br>Summary of<br>Free & Total<br>CCL17 in<br>Serum<br>Concentration-<br>Time Data<br>(pg/mL) | Please only present the median, min, max, sd (log), geometric mean and 95% CI back-transformed from the loge scale. Apply logit transformation for % reduction parameter. If % reduction ≤0, set to 0.1. If % reduction ≥100, set to 99.9. These imputations are needed for logit transformation. Use Student's t-distribution for CI. Please only present the median, min, max, sd (log), geometric mean and 95% CI back-transformed from the loge scale. Apply logit transformation for % reduction parameter and present median, min, max, sd (logit), geometric mean and 95% CI back-transformed from the logit scale. If % reduction ≤0, set to 0.1. If % reduction ≥100, set to 99.9. These imputations are needed for logit transformation. Use Student's t-distribution for CI. Add the following footnotes: Note: Free CCL17 values below the LLOQ have been imputed to ½*LLOQ. Total CCL17 values below the LLOQ whilst missing baseline values have been imputed to the median of the non-missing baseline values. Note: Free CCL17 and Total CCL17 exceeding the upper limit of quantification (ULOQ) have been excluded from the summary statistics (ULOQ Free CCL17: 3600 pg/mL, ULOQ Total CCL17: 50000 pg/mL). Note: If more than 30% of values have been imputed at any timepoint for a treatment group, then the standard deviation is not displayed. Note: Baseline is the mean of the Day -4 and Day 1 Pre-Dose assessments. Note: Percentage reduction and fold increase parameters were calculated using a model based post-hoc analysis. Note: Percentage reduction values <= 0 are imputed to be 0.1 and values >= 100 are imputed to be 99.9. | Part B SAC |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| | | | | Note: The percentage reduction parameter was logit transformed, summarised, and back-transformed using the logistic function to obtain the geometric summary statistics. The 95% CI of the geometric mean was calculated using Student's t distribution. | |
| | Safety | PD_T2 | Part B: Summary of Model-Derived Free and Total CCL17 in Serum Target Engagement Parameters (non- transformed and log- transformed) | Please only present the median, min, max, sd (log), geometric mean and 95% CI back-transformed from the loge scale. Please note that tmin and tmax should not be loge-transformed and 95% CI should not be presented. Apply logit transformation for % reduction and maximum % reduction parameters. If % reduction ≤0, set to 0.1. If % reduction ≥100, set to 99.9. These imputations are needed for logit transformation. Use Student's t-distribution for CI. Add the following footnotes: Note: All Target Engagement parameters were calculated using a model based posthoc analysis. Note: Percentage reduction values <= 0 are imputed to be 0.1 and values >= 100 are imputed to be 99.9. Note: The percentage reduction and maximum percentage reduction parameters were logit transformed, summarised, and back-transformed using the logistic function to obtain the geometric summary statistics. The 95% CI of the geometric mean was calculated using Student's t distribution. | IA3, Part B<br>SAC |
| Imm | unogenicity | | | | |
| 4.08. | Safety | IMM1 | Part B:<br>Summary of<br>Immunogenicity | Add extra row for Part B SAC - "Highest post-baseline" result. This would be #participants with at least one post-baseline positive result / # participants with at least one post baseline sample. | IA3, Part B<br>SAC |

# 14.11.11. Pharmacodynamic Figures

### 14.11.11.1. Part A

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Serum | n Target Engag | ement | | | |
| 4.01. | Safety | PK16 | Part A: Individual<br>Free & Total<br>Serum CCL17<br>Concentration-<br>Time Plots<br>(Linear and<br>Semi-log) | One panel per dose group. Add the following footnotes: Note: Free CCL17 LLOQ = 2.93 pg/mL, ULOQ = 3600 pg/mL. Note: Total CCL17 LLOQ = 13.11 pg/mL, ULOQ = 50000 pg/mL. Note: The baseline value is presented at an actual relative time of 0 days. Note: Any non-quantifiable (NQ) Free CCL17 concentration values have been set to ½*LLOQ. Note: Any NQ Total CCL17 concentration values before the first measurable concentration have been set to 0 and have been included in the linear plot. Note: Any single NQ values have been omitted. Note: Any multiple mid-profile NQ concentrations of Free CCL17 and Total CCL17 have been set to ½*LLOQ and 0, respectively, and the subsequent measurable concentrations have been retained. Note: Percentage reduction values <= 0 are imputed to be 0.1 and values >= 100 are imputed to be 99.9 | Part A SAC |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| 4.02. | Safety | PK17 | Part A: Mean<br>Free & Total<br>Serum CCL17<br>Concentration-<br>Time Plots<br>(Linear and<br>Semi-log) | Apply logit transformation for % reduction parameter. If % reduction ≤0, set to 0.1. If % reduction ≥100, set to 99.9. These imputations are needed for logit transformation. Use Student's t-distribution for Cl. Add the following footnotes: Note: Free CCL17 LLOQ = 2.93 pg/mL, ULOQ = 3600 pg/mL. Note: Total CCL17 LLOQ = 13.11 pg/mL, ULOQ = 50000 pg/mL. Note: Free CCL17 and Total CCL17 concentrations below LLOQ have been set to ½*LLOQ and 0, respectively, and have been included in the summary statistic calculations. Note: Any single mid-profile non-quantifiable (NQ) concentrations have been omitted. Note: Measurable Total CCL17 concentrations following more than one consecutive mid-profile NQ have been omitted. Note: Zero Total CCL17 concentration values have been set to missing in the log-linear plot. Note: The geometric mean is plotted as the data is not normally distributed. Note: Percentage reduction values <= 0 are imputed to be 0.1 and values >= 100 are imputed to be 99.9. Note: The percentage reduction parameter was logit transformed, summarised, and back-transformed using the logistic function to obtain the geometric summary statistics. | Part A SAC |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| 4.03. | Safety | PK18 | Part A: Median<br>Free & Total<br>Serum CCL17<br>Concentration-<br>Time Plots<br>(Linear and<br>Semi-log) | .Add the following footnotes: Note: Free CCL17 LLOQ = 2.93 pg/mL, ULOQ = 3600 pg/mL. Note: Total CCL17 LLOQ = 13.11 pg/mL, ULOQ = 50000 pg/mL. Note: Free CCL17 and Total CCL17 concentrations below LLOQ have been set to ½*LLOQ and 0, respectively, and have been included in the summary statistic calculations. Note: Any single mid-profile non-quantifiable (NQ) concentrations have been omitted. Note: Measurable Total CCL17 concentrations following more than one consecutive mid-profile NQ have been omitted. Note: Zero Total CCL17 concentration values have been set to missing in the log-linear plot. | Part A SAC |
### 14.11.11.2. Part B

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Serun | Target Engag | ement | | | |
| 4.04. | Safety | PK16 | Part B: Individual Free & Total Serum CCL17 Concentration-Time Plots (Linear and Semi-log) | One panel per dose group. Add the following footnotes: Note: Free CCL17 LLOQ = 2.93 pg/mL, ULOQ = 3600 pg/mL. Note: Total CCL17 LLOQ = 13.11 pg/mL, ULOQ = 50000 pg/mL. Note: The baseline value is presented at an actual relative time of 0 days. Note: Any non-quantifiable (NQ) Free CCL17 concentration values have been set to ½*LLOQ. Note: Any NQ Total CCL17 concentration values before the first measurable concentration have been set to 0 and have been included in the linear plot. Note: Any single NQ values have been omitted. Note: Any multiple mid-profile NQ concentrations of Free CCL17 and Total CCL17 have been set to ½*LLOQ and 0, respectively, and the subsequent measurable concentrations have been retained. Note: Percentage reduction values <= 0 are imputed to be 0.1 and values >= 100 are imputed to be 99.9. | Part B SAC |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| 4.05. | Safety | PK17 | Part B: Mean Free & Total<br>Serum CCL17<br>Concentration-Time Plots<br>(Linear and Semi-log) | Apply logit transformation for % reduction parameter. If % reduction ≤0, set to 0.1. If % reduction ≥100, set to 99.9. These imputations are needed for logit transformation. Use Student's t-distribution for CI. Add the following footnotes: Note: Free CCL17 LLOQ = 2.93 pg/mL, ULOQ = 3600 pg/mL. Note: Total CCL17 LLOQ = 13.11 pg/mL, ULOQ = 50000 pg/mL. Note: Free CCL17 and Total CCL17 concentrations below LLOQ have been set to ½*LLOQ and 0, respectively, and have been included in the summary statistic calculations. Note: Any single mid-profile non-quantifiable (NQ) concentrations have been omitted. Note: Measurable Total CCL17 concentrations following more than one consecutive mid-profile NQ have been omitted. Note: Zero Total CCL17 concentration values have been set to missing in the log-linear plot. Note: The geometric mean is plotted as the data is not normally distributed. Note: Percentage reduction values <= 0 are imputed to be 0.1 and values >= 100 are imputed to be 99.9. Note: The percentage reduction parameter was logit transformed, summarised, and back-transformed using the logistic function to obtain the geometric summary statistics. | Part B SAC |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| 4.06. | Safety | PK18 | Part B: Median Free & Total<br>Serum CCL17<br>Concentration-Time Plots<br>(Linear and Semi-log) | Add the following footnotes: Note: Free CCL17 LLOQ = 2.93 pg/mL, ULOQ = 3600 pg/mL. Note: Total CCL17 LLOQ = 13.11 pg/mL, ULOQ = 50000 pg/mL. Note: Free CCL17 and Total CCL17 concentrations below LLOQ have been set to ½*LLOQ and 0, respectively, and have been included in the summary statistic calculations. Note: Any single mid-profile non-quantifiable (NQ) concentrations have been omitted. Note: Measurable Total CCL17 concentrations following more than one consecutive mid-profile NQ have been omitted. Note: Zero Total CCL17-concentration values have been set to missing in the log-linear plot. | Part B SAC |

### 14.11.12. Biomarker Tables

### 14.11.12.1. Part A

| No. | Population | IDSL/<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Immur | e Cell Phenoty | /pe | | | |
| 5.01. | Biomarker | BIO_T1 | Part A: Summary of Immune Cell Phenotypes | | Part A SAC |
| 5.02. | Biomarker | BIO_T2 | Part A: Analyses of Immune Cell Phenotypes: Treatment | | Part A SAC |
| 5.03. | Biomarker | BIO_T3 | Part A: Analyses of Immune Cell Phenotypes: Sample Type | | Part A SAC |

# 14.11.13. Biomarker Figures

### 14.11.13.1. Part A

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Immur | ne Cell Phenoty | уре | | | |
| 5.01. | Biomarker | BIO_F1 | Part A: LS Mean Change from Baseline (+/- SE) of Immune Cell Phenotypes: Treatments by Visit | | Part A SAC |
| 5.02. | Biomarker | BIO_F2 | Part A: Differences and 95% CI of Immune Cell Phenotypes: Treatments by Visit | | Part A SAC |
| 5.03. | Biomarker | BIO_F1 | Part A: LS Mean Change from Baseline (+/- SE) of Immune Cell Phenotypes: Sample Type by Visit | | Part A SAC |
| 5.04. | Biomarker | BIO_F2 | Part A: Differences and 95% CI of Immune Cell Phenotypes: Sample Type by Visit | | Part A SAC |

# 14.11.14. Efficacy Tables

### 14.11.14.1. Part B

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Primary | Efficacy | | | | |
| 6.01. | ITT | EFF_T10 | Part B: Summary of Pain Intensity Data | Frequency table showing at each visit, how many subjects had how many days of knee pain intensity data (presented by trt group). | IA1, IA2,<br>Part B SAC |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 6.02. | ПТ | EFF_T1 | Part B: Summary of Absolute Values and Change from Baseline in Average Knee Pain Intensity | | IA1, IA2, IA3,<br>IA4,<br>Part B SAC |
| 6.03. | Ш | EFF_T2 | Part B: Bayesian Analysis of Change from Baseline in Average Knee Pain Intensity | | IA1, IA2, IA3,<br>IA4,<br>Part B SAC |
| 6.04. | PP | EFF_T1 | Part B: Summary of Absolute Values and Change from Baseline in Average Knee Pain Intensity | | Part B SAC |
| 6.05. | PP | EFF_T2 | Part B: Bayesian Analysis of Change from Baseline in<br>Average Knee Pain Intensity | | Part B SAC |
| 6.06. | ПТ | EFF_T1 | Part B: Summary of Absolute Values and Change from Baseline in Worst Knee Pain Intensity | | IA3, IA4, Part<br>B SAC |
| 6.07. | ΙΤΤ | EFF_T2 | Part B: Bayesian Analysis of Change from Baseline in Worst Knee Pain Intensity | | IA3, IA4, Part<br>B SAC |







# 14.11.15. Efficacy Figures

### 14.11.15.1. Part B

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Prima | ry Efficacy | | | | |
| 6.01. | Ш | EFF_F1 | Part B: Plot of Posterior Median and 95% CI of Average<br>Knee Pain Intensity | | Part B SAC |
| 6.02. | ш | EFF_F1 | Part B: Plot of Posterior Median and 95% CI of Change from Baseline in Average Knee Pain Intensity | | IA1, IA2, IA3,<br>IA4,<br>Part B SAC |
| 6.03. | IΠ | EFF_F1 | Part B: Plot of Posterior Median and 95% CI of Worst<br>Knee Pain Intensity | | Part B SAC |
| 6.04. | ш | EFF_F1 | Part B: Plot of Posterior Median and 95% CI of Change from Baseline in Worst Knee Pain Intensity | | Part B SAC |
| 6.05. | PP | EFF_F1 | Part B: Plot of Posterior Median and 95% CI of Average<br>Knee Pain Intensity | | Part B SAC |
| 6.06. | PP | EFF_F1 | Part B: Plot of Posterior Median and 95% CI of Change from Baseline in Average Knee Pain Intensity | | Part B SAC |



# 14.11.16. ICH Listings

### 14.11.16.1. Part A

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Subje | ct Disposition | 1 | | | |
| 1. | Screened | ES7 | Part A: Listing of Reasons for Screen Failure | | Part A SAC |
| 2. | Screened | ES9 | Part A: Listing of Subjects who were Rescreened | | Part A SAC |
| 3. | Enrolled | ES2 | Part A: Listing of Reasons for Study Withdrawal | | Part A SAC |
| 4. | Randomized | BL1 | Part A: Listing of Subjects for Whom the Treatment Blind was Broken | | Part A SAC |
| 5. | Randomized | TA1 | Part A: Listing of Planned and Actual Treatments | | Part A SAC |
| Proto | col Deviations | ·I | , | 1 | 1 |
| 6. | Enrolled | DV2 | Part A: Listing of Important Protocol Deviations | | Part A SAC |
| 7. | Enrolled | IE3 | Part A: Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | Part A SAC |
| Popul | ations Analysed | | | | |
| 8. | Enrolled | SP3 | Part A: Listing of Subjects Excluded from Any Population | | Part A SAC |
| Demo | graphic and Base | eline Charac | teristics | | |
| 9. | Randomized | DM2 | Part A: Listing of Demographic Characteristics | | Part A SAC |
| 10. | Randomized | DM9 | Part A: Listing of Race | | Part A SAC |
| Medic | al History | | | | |
| 11. | Safety | MH2 | Part A: Listing of Current and Past Medical Conditions | | Part A SAC |

| | | IDSL / | | | |
|---|---|---|---|---|---|
| No. | Population | Example Shell | Title | Programming Notes | Deliverable |
| Conc | omitant Medicati | ons | | | <u> </u> |
| 12. | Safety | CP_CM3 | Part A: Listing of Prior and Concomitant Medications | | Part A SAC |
| Expos | sure | | | | |
| 13. | Safety | POP_L01 | Part A: Listing of Exposure Data | | Part A SAC |
| Adve | se Events | | | | |
| 14. | Safety | AE8CP | Part A: Listing of All Adverse Events | | Part A SAC |
| 15. | Safety | AE7 | Part A: Listing of Subject Numbers for Individual Adverse Events | | Part A SAC |
| 16. | Safety | AE2 | Part A: Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | | Part A SAC |
| Serio | us and Other Sig | nificant Adv | erse Events | | |
| 17. | Safety | AE8CPa | Part A: Listing of Serious Adverse Events (Fatal and Non-Fatal) | | Part A SAC |
| 18. | Safety | AE14 | Part A: Listing of Reasons for Considering as a Serious Adverse Event | | Part A SAC |
| 19. | Safety | AE8CP | Part A: Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | | Part A SAC |
| 20. | Safety | AE8CP | Part A: Listing of Other Significant Adverse Events | | Part A SAC |
| Vital S | Signs | • | | | |
| 21. | Safety | VS4 | Part A: Listing of Vital Signs of Potential Clinical Importance | | Part A SAC |
| 22. | Safety | VS4 | Part A: Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance | | Part A SAC |
| Labor | atory: All | | | | <u> </u> |
| 23. | Safety | LB5 | Part A: Listing of Laboratory Values of Potential Clinical Importance | | Part A SAC |
| 24. | Safety | LB5 | Part A: Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance | | Part A SAC |
| 25. | Safety | LB14 | Part A: Listing of Laboratory Data with Character Results | | Part A SAC |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| 26. | Safety | UR2A | Part A: Listing of Urinalysis Data for Subjects with Any Value of Potential Clinical Importance | | Part A SAC |
| ECG | | | | | |
| 27. | Safety | EG3 | Part A: Listing of ECG Values of Potential Clinical Importance | | Part A SAC |
| 28. | Safety | EG3 | Part A: Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | | Part A SAC |
| 29. | Safety | EG5 | Part A: Listing of Abnormal ECG Findings | | Part A SAC |
| 30. | Safety | EG5 | Part A: Listing of All ECG Findings for Subjects with an Abnormal ECG Finding | | Part A SAC |
| Telem | elemetry | | | | |
| 31. | Safety | EG5 | Part A: Listing of Abnormal Telemetry Findings | | Part A SAC |

### 14.11.16.2. Part B

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Subjec | t Disposition | | | | |
| 32. | Screened | ES7 | Part B: Listing of Reasons for Screen Failures | | Part B SAC |
| 33. | Screened | ES9 | Part B: Listing of Subjects who were Rescreened | | Part B SAC |
| 34. | Enrolled | ES2 | Part B: Listing of Reasons for Study Withdrawal | | Part B SAC |
| 35. | Randomized | BL1 | Part B: Listing of Subjects for Whom the Treatment Blind was Broken | | Part B SAC |
| 36. | ITT | SD2 | Part B: Listing of Reasons for Study Treatment Discontinuation | | Part B SAC |
| 37. | Randomized | TA1 | Part B: Listing of Planned and Actual Treatments | | Part B SAC |
| Protoc | rotocol Deviations | | | | |
| 38. | Enrolled | DV2 | Part B: Listing of Important Protocol Deviations | | Part B SAC |

| No. | Population | IDSL /<br>Example | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| 39. | Enrolled | Shell<br>IE3 | Part B: Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | Part B SAC |
| Popul | ations Analysed | | | | |
| 40. | Enrolled | SP3 | Part B: Listing of Subjects Excluded from Any Population | | Part B SAC |
| Demo | graphic and Bas | eline Charac | | | |
| 41. | Randomized | DM2 | Part B: Listing of Demographic Characteristics | | Part B SAC |
| 42. | Randomized | DM9 | Part B: Listing of Race | | |
| Medic | al Conditions | • | | | |
| 43. | Safety MH2 Part B: Listing of Current and Past Medical Conditions | | | Part B SAC | |
| Conce | omitant Medication | ons | | | |
| 44. | Safety | CP_CM3 | Part B: Listing of Prior and Concomitant Medications | | Part B SAC |
| 45. | Safety | CP_CM3 | Part B: Listing of Prior and Concomitant Osteoarthritis Medications | OA con-meds are captured on a specific CRF page | Part B SAC |
| Expos | sure | | | | |
| 46. | Safety | EX3 | Part B: Listing of Exposure Data | Include number of injections received | Part B SAC |
| Adver | se Events | | | | <u> </u> |
| 47. | Safety | AE8CP | Part B: Listing of All Adverse Events | | Part B SAC |
| 48. | Safety | AE7 | Part B: Listing of Subject Numbers for Individual Adverse Events | | Part B SAC |
| 49. | Safety AE2 Part B: Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | | | Part B SAC | |
| Serio | us and Other Sig | nificant Adve | | | • |
| 50. | Safety | AE8CPa | Part B: Listing of Serious Adverse Events (Fatal and Non-Fatal) | | |
| 51. | Safety | AE14 | Part B: Listing of Reasons for Considering as a Serious Adverse Event | | |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| 52. | Safety | AE8CP | Part B: Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | | IA3, Part B<br>SAC |
| 53. | Safety | AE8CP | Part B: Listing of Other Significant Adverse Events | | Part B SAC |
| Vital S | Signs | | | | |
| 54. | Safety | VS4 | Part B: Listing of Vital Signs of Potential Clinical Importance | | Part B SAC |
| 55. | Safety | VS4 | Part B: Listing of All Vital Signs Data for Subjects with Any Value of Potential Clinical Importance | | Part B SAC |
| Labor | atory: All | | | | |
| 56. | Safety | LB5 | Part B: Listing of Laboratory Values of Potential Clinical Importance | g of Laboratory Values of Potential Clinical | |
| 57. | Safety | LB5 | Part B: Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance | | IA3, Part B<br>SAC |
| 58. | Safety | LB14 | Part B: Listing of Laboratory Data with Character Results | | Part B SAC |
| 59. | Safety | UR2A | Part B: Listing of Urinalysis Data for Subjects with Any Value of Potential Clinical Importance | | Part B SAC |
| ECG | | | | | |
| 60. | Safety | EG3 | Part B: Listing of ECG Values of Potential Clinical Importance | | Part B SAC |
| 61. | Safety | EG3 | Part B: Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | | Part B SAC |
| 62. | Safety | EG5 | Part B: Listing of Abnormal ECG Findings | | Part B SAC |
| 63. | Safety | EG5 | art B: Listing of All ECG Findings for Subjects with an bnormal ECG Finding | | Part B SAC |

# 14.11.17. ICH Conditional Listings

The following listings will only be produced if a liver event is observed within the trial.

### 14.11.17.1. Part A

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Hepat | Hepatobiliary (Liver) | | | | |
| 64. | Safety | MH2 | Part A: Listing of Medical Conditions for Subjects with | Conditional on liver event being | Part A SAC |
| 04. | Salety | IVII IZ | Liver Stopping Events | seen | T all A SAC |
| 65. | Safety | SU2 | Part A: Listing of Substance Use for Subjects with Liver | Conditional on liver event being | Part A SAC |
| 03. | Salety | 302 | Stopping Events | seen | rait A SAC |

### 14.11.17.2. Part B

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Hepat | Hepatobiliary (Liver) | | | | |
| 66. | Safety | afety MH2 | Part B: Listing of Medical Conditions for Subjects with | Conditional on liver event being | Part B SAC |
| 00. | Salety | IVII IZ | Liver Stopping Events | seen | Fall D SAC |
| 67 | '. Safety | MH2 Part B: Li | Part B: Listing of Substance Use for Subjects with Liver | Conditional on liver event being | Part B SAC |
| 67. | Salety | IVITZ | Stopping Events | seen | Pail D SAC |

### 14.11.18. Non-ICH Listings

### 14.11.18.1. Part A

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Subs | ubstance Use | | | | |
| 68. | Safety | SU2 | Part A: Listing of Substance Use | Include columns: Smoking history,<br>Currently Smoke, Last Smoked,<br>Drink Alcohol, Units per Week,<br>Currently using Illicit Drugs | Part A SAC |
| Phari | macokinetics | | | | |
| <b>69</b> . | PK | PK07 | Part A: Listing of Serum GSK3858279 Concentration-<br>Time Data (ng/mL) | | Part A SAC |
| 70. | PK | PK13 | Part A: Listing of Derived Serum GSK3858279<br>Pharmacokinetic Parameters | Add a footnote saying that NQ means non-quantifiable and LLQ=100 ng/mL | Part A SAC |
| CCI | | | | | |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Pharr | harmacodynamic | | | | |
| 72. | Safety | PK07 | Part A: Listing of Free & Total CCL17 in Serum Concentration-Time Data (pg/mL) | Including Percentage Inhibition/Fold Increase Add a footnote saying that NQ means non-quantifiable and Free CCL17 LLOQ=2.93 pg/mL and Total CCL17 LLOQ=13.11 pg/mL. | Part A SAC |
| 73. | Safety | PK13 | Part A: Listing of Derived Free CCL17 in Serum Target Engagement Parameters | | Part A SAC |
| 74. | Safety | PK13 | Part A: Listing of Derived Total CCL17 in Serum<br>Target Engagement Parameters | | Part A SAC |
| 75. | Blister | PK07 | Part A: Listing of Free & Total CCL17 in Blister Fluid Concentration-Time Data (pg/mL) | Including Blister/Serum Ratio | Part A SAC |
| 76. | Safety | IMM2 | Part A: Listing of Immunogenicity | | Part A SAC |
| Biom | arker | | | | |
| 77. | Biomarker | BIO_L1 | Part A: Listing of Immune Cell Phenotypes | | Part A SAC |

### 14.11.18.2. Part B

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Subst | Substance Use | | | | |
| 78. | Safety | SU2 | Part B: Listing of Substance Use | Include columns: Smoking history, Currently Smoke, Last Smoked, Drink Alcohol, Units per Week, Currently using Illicit Drugs | Part B SAC |

| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| Pharr | narmacokinetics | | | | |
| 79. | PK | PK07 | Part B: Listing of Serum GSK3858279 Concentration-Time Data (ng/mL) | Add a footnote saying that NQ means non-<br>quantifiable and LLOQ=100 ng/mL | Part B SAC |
| 80. | PK | PK13 | Part B: Listing of Model-Derived Serum GSK3858279 Pharmacokinetic Parameters | Add a footnote saying that "All Pharmacokinetic parameters were calculated using a model based post-hoc analysis". | Part B SAC |
| Pharr | nacodynamic | | | | |
| 81. | Safety | PK07 | Part B: Listing of Free & Total CCL17 in Serum Concentration-Time Data (pg/mL) | Add a footnote saying that LLOQ means lower limit of quantification and ULOQ means upper limit of quantification. LLOQ for free CCL17= 2.93 pg/mL. LLOQ for total CCL17= 13.11 pg/mL.ULOQ for free CCL17= 3600 pg/mL. ULOQ for total CCL17= 50000 pg/mL. | Part B SAC |
| 82. | Safety | PK13 | Part B: Listing of Derived Free CCL17 in Serum Target Engagement Parameters | Including Percentage Inhibition/Fold Increase. Add a footnote saying "All Target Engagement parameters were calculated using a model based post-hoc analysis.". | Part B SAC |
| 83. | Safety | PK13 | Part B: Listing of Derived Total CCL17 in Serum Target Engagement Parameters | Add a footnote saying "All Target Engagement parameters were calculated using a model based post-hoc analysis.". | Part B SAC |
| 84. | Safety | IMM2 | Part B: Listing of Immunogenicity | For IA3, include only participants with at least one positive confirmation assay result. | IA3, Part B<br>SAC |
| Prima | ary Efficacy | | | | |
| 85. | ITT | EFF_L01 | Part B: Listing of Average and Worst Knee Pain Intensity | Include the number of records which make up the average | IA1, IA2,<br>Part B SAC |

| | No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|---|
| CCI | | | | | | |
| | COVID | )-19 | | | | |
| | 88. | Randomized | PAN7 | Part B: Listing of All Subjects with Visits and<br>Assessments Impacted by COVID-19<br>Pandemic | | Part B SAC |